

Statistical Analysis Plan

Verona Pharma PROTOCOL No. RPL554-CO-301


# STATISTICAL ANALYSIS PLAN

RPL554-CO-301

A PHASE III RANDOMIZED, DOUBLE-BLIND, PLACEBO-CONTROLLED STUDY TO EVALUATE THE EFFICACY AND SAFETY OF ENSIFENTRINE OVER 24 WEEKS (WITH A 48-WEEK SAFETY SUBSET) IN PATIENTS WITH MODERATE TO SEVERE CHRONIC OBSTRUCTIVE PULMONARY DISEASE

VERSION NUMBER AND DATE: FINAL V1.0 02NOV2022





Statistical Analysis Plan




Upon review of this document, the undersigned approves this version of the Statistical Analysis Plan, authorizing that the content is acceptable for the reporting of this study.







Statistical Analysis Plan


# MODIFICATION HISTORY

| Unique<br>Identifier<br>for this<br>Version | Date of the<br>Document<br>Version | Author | Significant Changes from<br>Previous Authorized Version |
|---|---|---|---|
| 0.1 | 28JAN2021 | Ruth Woodfine | Not Applicable – First Version |
| 0.2 | 24AUG2022 | Maria Cristina<br>Mwandigha | Separated analyses for weeks 24 and 48 strata and updated based on updated 302 SAP |
| 1.0 | 31OCT2022 | Maria Cristina<br>Mwandigha | Major updates based on client<br>comments such as handling Russian<br>labs, analysis of other efficacy<br>endpoints, and additional efficacy<br>endpoints |





Statistical Analysis Plan


## **ABBREVIATIONS**

| AE | Adverse Event |
|---|---|
| ALT | Alanine Aminotransferase |
| ANCOVA | Analysis of Covariance |
| AST | Aspartate Aminotransferase |
| ATC | Anatomical Therapeutic Clinical Classification System |
| AUC <sub>0-t</sub> | Area Under the Curve over t hours |
| BDI | Baseline Dyspnea Index |
| BDR | Blinded Data Review |
| BMI | Body Mass Index |
| BPM | Beats Per Minute |
| COPD | Chronic Obstructive Pulmonary Disease |
| CRF | Case Report Form |
| DBL | Database Lock |
| DBP | Diastolic Blood Pressure |
| DMC | Data Monitoring Committee |
| ECG | Echocardiogram |
| ENR | All Patients Enrolled |
| EOS | End of Study |
| EQ-5D-5L | EuroQol-5-Domain Questionnaire |
| E-RS <sup>TM</sup> : COPD | Evaluating Respiratory Symptoms for COPD |
| ERT | eResearch Technology |
| FEV <sub>1</sub> | Forced Expiratory Volume in 1 second |
| FVC | Forced Vital Capacity |
| GGT | Gamma Glutamyltransferase |
| HRU | Healthcare Resource Utilization |
| IV | Intravenous |
| LABA | Long Acting Beta 2 Agonist |
| LAMA | Long Acting Muscarinic Antagonist |
| LOCF | Last Observation Carried Forward |
| MedDRA | Medical Dictionary for Regulatory Activities |
| MI | Multiple Imputation |
| mITT | Modified Intent-to-Treat |
| mMRC | Modified Medical Research Council |
| MMRM | Mixed Model for Repeated Measures |
| PD | Protocol Deviation |
| PP | Per-Protocol |
| PT | Preferred Term |





## Statistical Analysis Plan


| Qol | Quality of Life |
|------|-----------------------------------------------------------------|
| QTcF | QT interval corrected for heart rate using Fridericia's formula |
| RND | All Patients Randomized |
| SAP | Statistical Analysis Plan |
| SABA | Short Acting Beta 2 Agonist |
| SAE | Serious Adverse Event |
| SAF | Safety Analysis |
| SAS | Statistical Analysis Software |
| SBP | Systolic Blood Pressure |
| SD | Standard Deviation |
| SGRQ | St. George's Respiratory Questionnaire |
| SI | Standard International |
| SOC | System Organ Class |
| TDI | Transition Dyspnea Index |
| TEAE | Treatment-Emergent Adverse Event |
| WHO | World Health Organization |





Statistical Analysis Plan


# TABLE OF CONTENTS

| 1.<br>2. | STUDY OBJECTIVES AND ESTIMANDS | |
|---|---|---|
| 2.1. | Primary Objective | 12 |
| 2.2. | Secondary Objectives | 12 |
| 2.3. | Other Objectives | 12 |
| 2.4. | Safety Objectives | 12 |
| 2.5. | Estimands | 12 |
| 3. | STUDY DESIGN | 16 |
| 3.1. | General Description | 16 |
| 3.2. | Schedule of Events | 17 |
| 3.3. | Changes to Analysis from Protocol | 17 |
| 4. | PLANNED ANALYSES | 18 |
| 4.<br>4.1. | PLANNED ANALYSES Data Monitoring Committee (DMC) | |
| | | 18 |
| 4.1. | Data Monitoring Committee (DMC) | 18 |
| 4.1.<br>4.2. | Data Monitoring Committee (DMC) | 18<br>18 |
| 4.1.<br>4.2.<br>4.3. | Data Monitoring Committee (DMC) | 18 |
| 4.1.<br>4.2.<br>4.3. | Data Monitoring Committee (DMC) | 18 |
| 4.1.<br>4.2.<br>4.3.<br>5. | Data Monitoring Committee (DMC) | 18 |
| 4.1.<br>4.2.<br>4.3.<br>5.<br>5.1. | Data Monitoring Committee (DMC) | 1818182020 |



## Statistical Analysis Plan


| 5.7. Per-Protocol Population 2 5.8. Safety Analysis Set 2 5.9. Extended Safety Analysis Set 2 6. GENERAL CONSIDERATIONS 2 6.1. Reference Dates and Study Day 2 6.2. Baseline 2 6.3. Retests, Unscheduled Visits and Early Termination Data 2 6.4. Windowing Conventions 2 6.5. Statistical Tests 3 6.6. Common Calculations 3 6.7. Actual Treatment 3 6.8. Software Version 3 6.9. Strata Calculations 3 6.10. Russian Laboratories 3 7. STATISTICAL CONSIDERATIONS 3 7.1. Adjustments for Covariates and Factors to be Included in Analyses 3 7.2. Multicenter Studies 3 7.3. Missing data 3 7.4. Multiple Comparisons/ Multiplicity 3 7.5. Examination of Subgroups 3 8. OUTPUT PRESENTATIONS 3 9. DISPOSITION AND WITHDRAWALS 3 | 5.6. | Extended modified Intent-to-Treat Population | 20 |
|---|---|---|---|
| 5.9. Extended Safety Analysis Set 2 6. GENERAL CONSIDERATIONS 2 6.1. Reference Dates and Study Day 2 6.2. Baseline 2 6.3. Refests, Unscheduled Visits and Early Termination Data 2 6.4. Windowing Conventions 2 6.5. Statistical Tests 3 6.6. Common Calculations 3 6.7. Actual Treatment 3 6.8. Software Version 3 6.9. Strata Calculations 3 6.10. Russian Laboratories 3 7. STATISTICAL CONSIDERATIONS 3 7.1. Adjustments for Covariates and Factors to be Included in Analyses 3 7.2. Multicenter Studies 3 7.3. Missing data 3 7.4. Multiple Comparisons/ Multiplicity 3 7.5. Examination of Subgroups 3 8. OUTPUT PRESENTATIONS 3 | 5.7. | Per-Protocol Population | 21 |
| 6. GENERAL CONSIDERATIONS 2 6.1. Reference Dates and Study Day 2 6.2. Baseline 2 6.3. Retests, Unscheduled Visits and Early Termination Data 2 6.4. Windowing Conventions 2 6.5. Statistical Tests 3 6.6. Common Calculations 3 6.7. Actual Treatment 3 6.8. Software Version 3 6.9. Strata Calculations 3 6.10. Russian Laboratories 3 7. STATISTICAL CONSIDERATIONS 3 7.1. Adjustments for Covariates and Factors to be Included in Analyses 3 7.2. Multicenter Studies 3 7.3. Missing data 3 7.4. Multiple Comparisons/ Multiplicity 3 7.5. Examination of Subgroups 3 8. OUTPUT PRESENTATIONS 3 | 5.8. | Safety Analysis Set | 21 |
| 6.1. Reference Dates and Study Day 2 6.2. Baseline 2 6.3. Retests, Unscheduled Visits and Early Termination Data 2 6.4. Windowing Conventions 2 6.5. Statistical Tests 3 6.6. Common Calculations 3 6.7. Actual Treatment 3 6.8. Software Version 3 6.9. Strata Calculations 3 6.10. Russian Laboratories 3 7. STATISTICAL CONSIDERATIONS 3 7.1. Adjustments for Covariates and Factors to be Included in Analyses 3 7.2. Multicenter Studies 3 7.3. Missing data 3 7.4. Multiple Comparisons/ Multiplicity 3 7.5. Examination of Subgroups 3 8. OUTPUT PRESENTATIONS 3 | 5.9. | Extended Safety Analysis Set | 21 |
| 6.2. Baseline 2 6.3. Retests, Unscheduled Visits and Early Termination Data 2 6.4. Windowing Conventions 2 6.5. Statistical Tests 3 6.6. Common Calculations 3 6.7. Actual Treatment 3 6.8. Software Version 3 6.9. Strata Calculations 3 6.10. Russian Laboratories 3 7. STATISTICAL CONSIDERATIONS 3 7.1. Adjustments for Covariates and Factors to be Included in Analyses 3 7.2. Multicenter Studies 3 7.3. Missing data 3 7.4. Multiple Comparisons/ Multiplicity 3 7.5. Examination of Subgroups 3 8. OUTPUT PRESENTATIONS 3 | 6. | GENERAL CONSIDERATIONS | 22 |
| 6.3. Retests, Unscheduled Visits and Early Termination Data 2 6.4. Windowing Conventions 2 6.5. Statistical Tests 3 6.6. Common Calculations 3 6.7. Actual Treatment 3 6.8. Software Version 3 6.9. Strata Calculations 3 6.10. Russian Laboratories 3 7. STATISTICAL CONSIDERATIONS 3 7.1. Adjustments for Covariates and Factors to be Included in Analyses 3 7.2. Multicenter Studies 3 7.3. Missing data 3 7.4. Multiple Comparisons/ Multiplicity 3 7.5. Examination of Subgroups 3 8. OUTPUT PRESENTATIONS 3 | 6.1. | Reference Dates and Study Day | 22 |
| 6.4. Windowing Conventions 2 6.5. Statistical Tests 3 6.6. Common Calculations 3 6.7. Actual Treatment 3 6.8. Software Version 3 6.9. Strata Calculations 3 6.10. Russian Laboratories 3 7. STATISTICAL CONSIDERATIONS 3 7.1. Adjustments for Covariates and Factors to be Included in Analyses 3 7.2. Multicenter Studies 3 7.3. Missing data 3 7.4. Multiple Comparisons/ Multiplicity 3 7.5. Examination of Subgroups 3 8. OUTPUT PRESENTATIONS 3 | 6.2. | Baseline | 22 |
| 6.5. Statistical Tests 3 6.6. Common Calculations 3 6.7. Actual Treatment 3 6.8. Software Version 3 6.9. Strata Calculations 3 6.10. Russian Laboratories 3 7. STATISTICAL CONSIDERATIONS 3 7.1. Adjustments for Covariates and Factors to be Included in Analyses 3 7.2. Multicenter Studies 3 7.3. Missing data 3 7.4. Multiple Comparisons/ Multiplicity 3 7.5. Examination of Subgroups 3 8. OUTPUT PRESENTATIONS 3 | 6.3. | Retests, Unscheduled Visits and Early Termination Data | 23 |
| 6.6. Common Calculations 3 6.7. Actual Treatment 3 6.8. Software Version 3 6.9. Strata Calculations 3 6.10. Russian Laboratories 3 7. STATISTICAL CONSIDERATIONS 3 7.1. Adjustments for Covariates and Factors to be Included in Analyses 3 7.2. Multicenter Studies 3 7.3. Missing data 3 7.4. Multiple Comparisons/ Multiplicity 3 7.5. Examination of Subgroups 3 8. OUTPUT PRESENTATIONS 3 | 6.4. | Windowing Conventions | 23 |
| 6.7. Actual Treatment 3 6.8. Software Version 3 6.9. Strata Calculations 3 6.10. Russian Laboratories 3 7. STATISTICAL CONSIDERATIONS 3 7.1. Adjustments for Covariates and Factors to be Included in Analyses 3 7.2. Multicenter Studies 3 7.3. Missing data 3 7.4. Multiple Comparisons/ Multiplicity 3 7.5. Examination of Subgroups 3 8. OUTPUT PRESENTATIONS 3 | 6.5. | Statistical Tests | 30 |
| 6.8. Software Version | 6.6. | Common Calculations | 30 |
| 6.9. Strata Calculations 3 6.10. Russian Laboratories 3 7. STATISTICAL CONSIDERATIONS 3 7.1. Adjustments for Covariates and Factors to be Included in Analyses 3 7.2. Multicenter Studies 3 7.3. Missing data 3 7.4. Multiple Comparisons/ Multiplicity 3 7.5. Examination of Subgroups 3 8. OUTPUT PRESENTATIONS 3 | 6.7. | Actual Treatment | 30 |
| 6.10. Russian Laboratories | 6.8. | Software Version | 31 |
| 7. STATISTICAL CONSIDERATIONS | 6.9. | Strata Calculations | 31 |
| 7.1. Adjustments for Covariates and Factors to be Included in Analyses | 6.10. | Russian Laboratories | 31 |
| 7.2. Multicenter Studies | 7. | STATISTICAL CONSIDERATIONS | 32 |
| 7.3. Missing data | 7.1. | Adjustments for Covariates and Factors to be Included in Analyses | 32 |
| 7.4. Multiple Comparisons/ Multiplicity | 7.2. | Multicenter Studies | 32 |
| 7.5. Examination of Subgroups | 7.3. | Missing data | 33 |
| 8. OUTPUT PRESENTATIONS | 7.4. | Multiple Comparisons/ Multiplicity | 33 |
| | 7.5. | Examination of Subgroups | 33 |



| Statistical | Analy | vsis | Plan |
|-------------|----------|-------|--------|
| Clationical | / VIIIGI | y 313 | I IGII |


| 9.2. Protocol Deviations | 37 |
|----------------------------------------------------|-------------------------|
| 9.3. Evaluation including excluded sites | 37 |
| 10. DEMOGRAPHIC AND OTHER BASI | ELINE CHARACTERISTICS37 |
| 10.1. Derivations | 38 |
| 10.2. Evaluation including excluded sites | 38 |
| | XY39 |
| 14. STUDY MEDICATION EXPOSURE | 41 |
| 14.1. Derivations | 41 |
| 15. COMPLIANCE | 41 |
| 15.1. Study Medication Compliance | 41 |
| 15.2. E-diary compliance | 44 |
| | 44 |
| 16. EFFICACY OUTCOMES | 45 |
| | 45 |
| | Variable |
| | le |
| | iable |
| 16.2. Secondary Efficacy | 49 |
| 16.2.1. Secondary Efficacy Variables & Derivations | 49 |
| | 52 y variables |




| Statistical Analysis Plan |
|---------------------------|

| 16222 | 207 - 4 - 1 - 1 - 1 - 1 - 1 - 1 | - |
|---|---|---|
| 16.2.2.2. | MI method – binary data | |
| 16.2.2.3. | MI method – range data | |
| 16.2.2.4. | Other methods | |
| | alysis of Secondary Efficacy Variables | |
| 16.2.3.1. | Change from baseline variables, incl. TDI | |
| 16.2.3.2. | Proportion of SGRQ total responders | |
| 16.2.4. Ser | sitivity Analysis of Secondary Efficacy Variables | 50 |
| 16.3. Othe | r Efficacy | 5 |
| | ner Efficacy Variables & Derivations | |
| 16.3.1.1. | COPD exacerbation | |
| 16.3.1.2. | Time to study withdrawal | |
| 16.3.1.3. | EQ-5D-5L | |
| 16.3.1.4. | HRU | |
| 16.3.1.5. | Patient Perception Survey | |
| 16.3.1.6. | | |
| 16.3.1.7. | FEV1 AUC <sub>6-12h</sub> | |
| | E-RS total score responder. | |
| 16.3.1.8. | Morning trough FEV <sub>1</sub> responder | |
| 16.3.1.9. | SGRQ domains | |
| 16.3.1.10. | | |
| | ssing Data Methods for Other Efficacy Variables | |
| | alysis of Other Efficacy Variables | |
| 16.3.4. Se | sitivity Analysis of Other Efficacy Variables | 62 |
| 16.4. Eval | nation including excluded sites | 62 |
| 16.4. Eval | nation including excluded sites | 62 |
| | TY OUTCOMES | |
| 17. SAFE | TY OUTCOMES | 63 |
| 17. SAFE | TY OUTCOMESrse Events | 63 |
| 17. SAFE 17.1. Adve | TY OUTCOMESrse Events | 63<br>65 |
| 17. SAFE 17.1. Adve 17.1.1. All 17.1.1.1. | TY OUTCOMES | |
| 17.1. Adve<br>17.1.1. Ali<br>17.1.1.1.<br>17.1.1.2. | TY OUTCOMES | |
| 17. SAFE 17.1. Adve 17.1.1. All 17.1.1.1. 17.1.1.2. 17.1.2. TE | TY OUTCOMES rse Events TEAEs Severity Relationship to Study Medication AEs Leading to Discontinuation of Study Medication | |
| 17. SAFE 17.1. Adve 17.1.1. 17.1.1.1. 17.1.1.2. TE 17.1.3. See | TY OUTCOMES rse Events TEAEs Severity Relationship to Study Medication AEs Leading to Discontinuation of Study Medication ious Adverse Events | |
| 17. SAFE 17.1. Adve 17.1.1. 17.1.1.1. 17.1.1.2. TE 17.1.3. See | TY OUTCOMES rse Events TEAEs Severity Relationship to Study Medication AEs Leading to Discontinuation of Study Medication | |
| 17. SAFE 17.1. Adve 17.1.1. All 17.1.1.2. 17.1.2. TE 17.1.3. Se 17.1.4. Ad | TY OUTCOMES rse Events TEAEs Severity Relationship to Study Medication AEs Leading to Discontinuation of Study Medication ious Adverse Events | |
| 17. SAFE 17.1. Adve 17.1.1. All 17.1.1.2. 17.1.2. TE 17.1.3. Se: 17.1.4. Ad 17.2. Labo | TY OUTCOMES | |
| 17. SAFE 17.1. Adve 17.1.1. All 17.1.1.1. 17.1.1.2. 17.1.2. TE 17.1.3. See 17.1.4. Ad 17.2. Labo 17.2.1. Lab | TY OUTCOMES | |
| 17. SAFE 17.1. Adve 17.1.1. All 17.1.1.1. 17.1.1.2. 17.1.2. TE 17.1.3. See 17.1.4. Ad 17.2. Labo 17.2.1. Lai 17.3. ECG | TY OUTCOMES | |
| 17. SAFE 17.1. Adve 17.1.1. All 17.1.1.1. 17.1.1.2. 17.1.2. TE 17.1.3. See 17.1.4. Ad 17.2. Labo 17.2.1. Lai 17.3. ECG | TY OUTCOMES | |
| 17. SAFE 17.1. Adve 17.1.1. All 17.1.1.1. 17.1.1.2. TE 17.1.3. Ser 17.1.4. Ad 17.2. Labo 17.2.1. La 17.3. ECG 17.3.1. ECG 17.4. Vital | rse Events TEAEs | |
| 17. SAFE 17.1. Adve 17.1.1. All 17.1.1.1. 17.1.1.2. TE 17.1.3. Ser 17.1.4. Ad 17.2. Labo 17.2.1. La 17.3. ECG 17.3.1. ECG 17.4. Vital | rse Events TEAEs | |
| 17. SAFE 17.1. Adve 17.1.1. All 17.1.1.1. 17.1.1.2. TE 17.1.3. Set 17.1.4. Add 17.2. Labo 17.2.1. Lai 17.3. ECG 17.3.1. ECG 17.4. Vital 17.4.1. Vital | rse Events TEAEs | |



| Statistical | Analy | ysis | Plan |
|-------------|-------|------|------|


| 17.6. Pneumonia | 70 |
|---|---|
| 17.7. Evaluation including excluded sites | 70 |
| 18. DATA NOT SUMMARIZED OR PRESENTED | 70 |
| 19. REFERENCES | |
| APPENDIX 1. PROGRAMMING CONVENTIONS FOR OUTPUTS | 72 |
| Dates & Times | 72 |
| Spelling Format | 72 |
| Presentation of Treatment Groups | 72 |
| Decimal Places | 72 |
| Presentation of Visits | 73 |
| Listings | 73 |
| Tables | 74 |
| APPENDIX 2. PARTIAL DATE CONVENTIONS | 75 |
| Algorithm for Treatment Emergence of Adverse Events: | 75 |
| Algorithm for Prior / Prior Concomitant / Concomitant Medications: | 76 |
| Algorithm for Concomitant Illnesses: | 79 |
| APPENDIX 3. ANNOTATED EXACT FOR RAW SCORE ASSIGNMENTAPPENDIX 4. RAW SUMMED SCORE TO SCALE CONVERSION TABLE FOR | 81 |
| EXACT TOTAL SCORE | 83 |
| APPENDIX 5. SGRQ ITEM WEIGHTS | 84 |
| APPENDIX 6. EQ-5D-5L WEIGHTS | 89 |
| Poland | 89 |
| England | 91 |
| US | 92 |





Statistical Analysis Plan


## 1. Introduction

This document describes the rules and conventions to be used in the presentation and analysis of efficacy and safety data for Protocol RPL554-CO-301. It describes the data to be summarized and analyzed, including specifics of the statistical analyses to be performed.

This statistical analysis plan (SAP) is based on protocol version 6.0, dated 18 February 2022.

A separate pooled SAP will be created which will include the details of pooled analysis between RPL554-CO-301 and RPL554-CO-302.

There will also be a separate blinded data review (BDR) plan that will outline the process for identification and decision making on patient's exclusion from analysis sets and on major protocol deviations. These will then be summarized in BDR report created for the data review outputs. This document will summarize each analysis set and reasons for the exclusion. In the BDR report protocol deviations (PDs) will also be outlined, specifying which patients were identified with each PD and whether these led to exclusion from the PP population. All analysis sets will be defined, and all possible PDs will be identified prior to unblinding.





Statistical Analysis Plan


## 2. STUDY OBJECTIVES AND ESTIMANDS

#### 2.1. PRIMARY OBJECTIVE

The primary objective of this study is to evaluate the efficacy of ensifentrine on lung function compared to placebo over a 12-hour dosing interval in patients with moderate to severe chronic obstructive pulmonary disease (COPD).

#### 2.2. SECONDARY OBJECTIVES

- To evaluate the effect of ensifentrine on other lung function parameters.
- To evaluate the effect of ensifentrine on COPD symptoms.
- To evaluate the effect of ensifentrine on health-related quality of life.

#### 2.3. OTHER OBJECTIVES

- To evaluate the effect of ensifentrine on moderate/severe COPD exacerbations.
- To evaluate the effect of ensifentrine on health utility and healthcare resource utilization (HRU).

#### 2.4. SAFETY OBJECTIVES

To evaluate the safety and tolerability of ensifentrine over 24 and 48 Weeks.

## 2.5. ESTIMANDS

The primary and secondary estimands to support regulatory decisions are described in Table 1.




Statistical Analysis Plan

List of Estimands Table 1;

| | | Attributes | | | |
|---|---|---|---|---|---|
| Estimand | Definition | Population | Variable/ Endpoint | Intercurrent event<br>handling strategy | Population-level summary measure |
| Primary | The efficacy of ensifentrine on lung function compared to placebo over a 12-hour dosing interval in patients with moderate to severe COPD. To evaluate the effect of ensifentrine on other lung function parameters. | Patients with moderate to severe COPD aged 40-80 years (inclusive) that are in the modified intent-to-treat (mITT) population. See full list of inclusion and exclusion criteria in Sections 5.1, 5.2 and 5.3 of study protocol. Patients with moderate to severe COPD aged 40-80 years (inclusive) that are in the mITT population. See full list of inclusion and exclusion criteria in Sections 5.1, 5.2 and 5.3 of study protocol. | Change from baseline forced expiratory volume in 1 second (FEV <sub>1</sub> ) to average FEV <sub>1</sub> area under the curve over 12 hours (AUC <sub>0-12h</sub> ) at Week 12. 1. Change from baseline FEV <sub>1</sub> to average FEV <sub>1</sub> AUC <sub>0-4h</sub> at Week 12. 2. Change from baseline FEV <sub>1</sub> to peak FEV <sub>1</sub> at Week 12. 3. Change from baseline FEV <sub>1</sub> to morning trough FEV <sub>1</sub> at Week | Regardless of whether the patient discontinues treatment prematurely and regardless of major protocol deviation, as per the Treatment Policy strategy. Regardless of whether the patient discontinues treatment prematurely and regardless of major protocol deviation, as per the Treatment Policy | Estimated treatment difference at Week 12 of the double-blind period (and corresponding 95% confidence interval [CI]) from analysis of covariance (ANCOVA) analysis. Estimated treatment difference at Week 12 of the double-blind period (and corresponding 95% CI) from ANCOVA analysis. |
| | | | 12 | strategy. | |



Copyright © 2009, 2010, 2012, 2016, 2018, 2019 IQVIA. All rights reserved. The contents of this document are confidential and proprietary to IQVIA Holdings Inc. and its subsidiaries. Unauthorized use, disclosure or reproduction is strictly prohibited.


Statistical Analysis Plan

| Estimated treatment difference at the end of the double-blind period (and corresponding 95% CI) from ANCOVA analysis. | 1. Estimated treatment difference at the end of the double-blind period (and corresponding 95% CI) from ANCOVA analysis. 2. Odds ratio for proportion of responders with an improvement of at least 4 units at the end of the double-blind period (and corresponding 95% CI) from logistic |
|---|---|
| Regardless of whether the patient discontinues treatment prematurely and regardless of major protocol deviation, as per the Treatment Policy strategy. | Regardless of whether the patient discontinues treatment prematurely and regardless of major protocol deviation, as per the Treatment Policy strategy. |
| Change from baseline (i.e. mean over the last 7 days of run-in) to the mean weekly value at Week 24 in COPD symptoms, as measured by daily diary (Evaluating Respiratory Symptoms for COPD [E-RS <sup>TM</sup> :COPD]) | Change from baseline in the St. George's Respiratory Questionnaire (SGRQ) total score at Week 24 Proportion of SGRQ responders at Week 24 |
| Patients with moderate to severe COPD aged 40-80 years (inclusive) that are in the mITT population. See full list of inclusion and exclusion criteria in Sections 5.1, 5.2 and 5.3 of study protocol. | Patients with moderate to severe COPD aged 40-80 years (inclusive) that are in the mITT population. See full list of inclusion and exclusion criteria in Sections 5.1, 5.2 and 5.3 of study protocol. |
| To evaluate the effect of ensifentrine on COPD symptoms. | To evaluate the effect of ensifentrine on health-related quality of life. |
| Secondary | Secondary |

Copyright © 2009, 2010, 2012, 2016, 2018, 2019 IQVIA. All rights reserved. The contents of this document are confidential and proprietary to IQVIA Holdings Inc. and its subsidiaries. Unauthorized use, disclosure or reproduction is strictly prohibited.



Statistical Analysis Plan

Verona Pharma PROTOCOL No. RPL554-CO-301

RPL554-CO-501

| regression analysis. |
|----------------------|



Copyright © 2009, 2010, 2012, 2016, 2018, 2019 IQVIA. All rights reserved. The contents of this document are confidential and proprietary to IQVIA Holdings Inc. and its subsidiaries. Unauthorized use, disclosure or reproduction is strictly prohibited.



Statistical Analysis Plan


## 3. STUDY DESIGN

#### 3.1. GENERAL DESCRIPTION

This is a Phase III, multicenter, randomized, double-blind, parallel group, placebo-controlled study. A flow chart illustrating the key components of the study is provided in Figure 1:

Figure 1: Study Flow Chart



Approximately 800 patients with moderate to severe COPD aged 40 to 80 years (inclusive) will be stratified by three different factors: treatment duration (48 or 24 weeks), stable background maintenance long-acting muscarinic antagonist (LAMA) or long-acting beta-2 agonist (LABA) monotherapy use (yes or no) and cigarette smoking (current or former). The 48-week stratum will be randomized 3:1 to receive ensifentrine (3 mg):placebo, and the 24-week stratum will be randomized 1:1 to receive ensifentrine (3 mg):placebo. Patients in the background maintenance LAMA or LABA therapy strata must withhold twice-daily maintenance LAMA or LABA (or LAMA/ICS or LABA/ICS) for 24 hours and once-daily maintenance LAMA or LABA (or LAMA/ICS or LABA/ICS) for 48 hours prior to initiation of any spirometry. All patients must withhold short acting beta-2 agonist (SABA) rescue medication for at least 4 hours prior to initiation of any spirometry.





Statistical Analysis Plan


Patients are expected to take the study medication twice daily, administered via a standard jet nebulizer, during the study period. Schedule of in-clinic dosing can be found in Section 1.4 of the study protocol.

#### 3.2. SCHEDULE OF EVENTS

Schedule of activities can be found in Section 1.3 of the study protocol.

## 3.3. CHANGES TO ANALYSIS FROM PROTOCOL

Changes to analysis from protocol include:

- · "COPD severity" added as a subgroup analysis.
- Sections 9.4.1 and 9.4.4 in the protocol states, "A sensitivity analysis [on the proportion of responders on the SGRQ] will be performed in which patients with missing data at the required visit will be considered non-responder in the analysis", and "For the responder analysis of SGRQ, patients with no available data for imputation will be considered non-responders as a sensitivity analysis", respectively. However, a non-responder analysis may create an unintentional bias in favor of the treatment arm, i.e. if placebo patients discontinue, this technique may inadvertently set more values in the placebo arm to "non-responder". Therefore, this technique for missing data analysis will not be implemented.
- Analysis of E-RS total score responder, defined as a decrease from baseline in the week mean total of E-RS score of greater than or equal to 2, added in the Section 16.3.1.6.
- Analysis of Morning trough FEV<sub>1</sub> responder, defined as an improvement from baseline of 100 mL or more, added in Section 16.3.1.7.
- Chronicity section removed from Adverse Event section.
- A sensitivity analysis will be performed for weekly mean E-RS total score, using ANCOVA approach, as described in Section  of the SAP, in which all patients with baseline mean = 0 will be excluded.
- Due to unreliability of the data, sites will be removed from efficacy and safety analyses in any section.
- Extended mITT and extended Safety populations set will be included as new populations to manage these sites being removed. Added in Section 5.
- Additional efficacy analysis of SGRQ and E-RS per domain using mITT population: SGRQ domains: Symptoms items 1 to 8; Activity items 11 and 15; Impacts items 9, 10, 12, 13, 14, 16 and 17 and E-RS domains: Breathlessness items 7, 8, 9, 10 and 11 (score range: 0-17); Cough and Sputum items 2, 3 and 4 (score range: 0-11); Chest Symptoms items 1, 5 and 6 (score range: 0-12)



Statistical Analysis Plan


## 4. PLANNED ANALYSES

A final analysis after database lock (DBL) is planned for this study.

## 4.1. DATA MONITORING COMMITTEE (DMC)

There will be no DMC for this study.

## 4.2. INTERIM ANALYSIS

There is no interim analysis planned for this study, however additional patients may be randomized if:

- the SD has increased significantly from the estimated 250 mL, as per sponsor discretion, and/or
- the withdrawal rate at 24 weeks exceeds 25% overall, and the percentage of patients with missing FEV<sub>1</sub> over 12 hours at Week 12 in mITT (modified Intent-to-Treat) population exceeds 20% overall.

Note: As part of the primary endpoint analysis, SD of the treatment difference is calculated to check the sample size with 90% power.

## 4.3. FINAL ANALYSIS

All final, planned analyses identified in this SAP will be performed by IQVIA Biostatistics following sponsor authorization of SAP (and associated output shells), DBL, analysis sets and unblinding of treatment.

## 5. ANALYSIS SETS

Agreement and authorization of patients included/excluded from each analysis set will be conducted prior to the unblinding of the study.

Analyses will be performed for the analysis sets described in Table 2.





Statistical Analysis Plan 

Table 2: Analysis sets

| | All<br>Patient<br>s<br>Enrolle<br>d Set | All<br>Patients<br>Rando<br>m. Set | Extende<br>d<br>Random<br>. Set | Modifie<br>d<br>Intent-<br>to-Treat<br>Pop. | Extende<br>d<br>modifie<br>d Intent-<br>to-Treat<br>Pop. | Per-<br>Protoc<br>ol Pop. | Safet<br>y Set | Extende<br>d Safety<br>Set |
|---|---|---|---|---|---|---|---|---|
| Disposition of patients | X | X | X | | | | | |
| Protocol<br>deviations | | X | | | | | | |
| Demographi<br>c and other<br>baseline<br>characteristi<br>cs | | X | X | X | X | | | |
| Surgical and<br>medical<br>history | | | | | | | X | |
| Prior and concomitant medication | | | | | | | X | |
| Compliance | | | | | | | X | |
| Efficacy:<br>Primary<br>endpoint | | | | X | X | X | | |
| Efficacy:<br>Secondary<br>endpoint | | | | X | X | X | | |
| Efficacy:<br>Other<br>endpoints | | | | X | | | | |
| Sensitivity<br>Analyses | | | | X | X | X | | |
| Safety | | | | | | | X | X |



Statistical Analysis Plan


## 5.1. PROCESS FOR ANALYSIS SET ASSIGNMENT

Analysis set assignments and any associated reasons for analyses set exclusion will be described in the BDR plan and finalized within the BDR report prior to unblinding.

## 5.2. ALL PATIENTS ENROLLED SET

The all patients enrolled (ENR) set will contain all patients who provide informed consent for this study. Patients will be classified according to randomized treatment with patients not randomized presented in a separate category, see Appendix 1. All patients enrolled will be summarized with and without subjects consented at sites

#### 5.3. ALL PATIENTS RANDOMIZED SET

The all patients randomized (RND) set will contain all patients in the ENR set who were randomized to study medication. For analyses and displays based on RND, patients will be classified according to randomized treatment. Sites number will be excluded from this population.

#### 5.4. EXTENDED RANDOMIZED SET

The Extended RND set will contain all patients in the ENR set who were randomized to study medication. For analyses and displays based on RND, patients will be classified according to randomized treatment. Sites number will be included in this population.

## 5.5. MODIFIED INTENT-TO-TREAT POPULATION

The mITT population will contain all patients in the RND set who received at least one dose (or partial dose) of study medication and patients will be classified according to randomized treatment. The intent-to-treat principle is preserved, despite the exclusion of patients randomized who did not take the study medication, because the decision of whether or not to begin the treatment could not be influenced by knowledge of the assigned treatment, i.e. the study medication is blinded. Sites number will be excluded from this population.

## 5.6. EXTENDED MODIFIED INTENT-TO-TREAT POPULATION

The Extended mITT population will contain all patients in the RND set who received at least one dose (or partial dose) of study medication and patients will be classified according to randomized treatment. The intent-to-treat principle is preserved, despite the exclusion of patients randomized





Statistical Analysis Plan


who did not take the study medication, because the decision of whether or not to begin the treatment could not be influenced by knowledge of the assigned treatment, i.e. the study medication is blinded. Sites number will be included in this population.

## 5.7. PER-PROTOCOL POPULATION

The per-protocol (PP) population will contain all patients in the mITT who did not discontinue the study medication before study day 74 and did not experience any major/important PDs considered to have an impact on efficacy assessments involving lung function at week 12. Reasons for exclusion will be specified at a BDR meeting prior to DBL and may include violations of inclusion/exclusion criteria, violations of withdrawal criteria, incorrect randomization, use of prohibited medication, did not follow blinding procedures and non-compliance. Patients will be classified according to randomized treatment. If protocol deviations in terms of dosing errors are detected post unblinding, these will lead to exclusion only if patient has received and used the opposite study drug compared to what was specified in the randomization and that this use occurred prior to week 12.

Patients who were excluded from PP due to the study medication being discontinued before study day 74 are not considered as protocol violations.

#### 5.8. SAFETY ANALYSIS SET

The safety analysis (SAF) set will contain all patients in the RND set who receive at least one dose (or partial dose) of study medication and patients will be classified according to treatment received.

If there is any doubt whether a patient was treated or not, they will be assumed treated for the purposes of analysis. Sites number will be excluded from this population.

#### 5.9. EXTENDED SAFETY ANALYSIS SET

The Extended SAF set will contain all patients in the RND set who receive at least one dose (or partial dose) of study medication and patients will be classified according to treatment received.

If there is any doubt whether a patient was treated or not, they will be assumed treated for the purposes of analysis. Sites number will be included in this population.



Copyright © 2009, 2010, 2012, 2016, 2018, 2019 IQVIA. All rights reserved. The contents of this document are confidential and proprietary to IQVIA Holdings Inc. and its subsidiaries. Unauthorized use, disclosure or reproduction is strictly prohibited.

Statistical Analysis Plan


## 6. GENERAL CONSIDERATIONS

## 6.1. REFERENCE DATES AND STUDY DAY

Study Day will be calculated from the reference start date and will be used to show start/stop day of assessments and events.

Reference start date is defined as the day of the first dose of study medication (Day 1 is the day of the first dose of study medication) and will appear in every listing where an assessment date or event date appears.

- If the date of the event is on or after the reference start date, then: Study Day = (date of event – reference start date) + 1.
- If the date of the event is prior to the reference start date, then: Study Day = (date of event – reference start date).

In the situation where the event date is partial or missing, the date will appear partial or missing in the listings, and Study Day, and any corresponding durations will be presented based on the imputations specified in Appendix 2 of the SAP.

Reference end date is defined as the date of the last dose of study medication.

#### 6.2. BASELINE

Unless otherwise specified, baseline is defined as the last non-missing measurement taken prior to reference start date (including unscheduled assessments). In the case where the last non-missing measurement and the reference start date coincide, that measurement will be considered baseline, unless time is present. If time of the assessment is on or after the study treatment start date, then the assessment is not considered baseline except in the following case: for main and responder SGRQ analysis, if the assessment on the day of randomization is done after dosing but prior to leaving the clinic after the 4 hour spirometry, the assessment is considered baseline. Adverse Events (AEs) and medications commencing on the reference start date will be considered post-baseline, ECG abnormalities from pre-dose assessments and laboratory abnormalities from pre-dose draws that are analyzed externally post-dose are still considered baseline.

Baseline for the spirometry endpoints is defined as the mean of the 2 measurements taken predose on Day 1 prior to reference start date and time, unless only 1 measurement is taken pre-dose on Day 1 prior to reference start date and time.





Statistical Analysis Plan


If the baseline visit is split across in 2 days with pre-dose assessments on Day -1 and dosing on Day 1, then measurement from day - 1 will constitute baseline for spirometry endpoints.

## 6.3. RETESTS, UNSCHEDULED VISITS AND EARLY TERMINATION DATA

In general, for by-visit summaries, data recorded at the nominal visit will be presented.

Patients who were a screen failure and received approval from the Medical Monitor for rescreening will go through all of the original screening assessments. Data from the latest rescreened visit will be used in the summaries, however all screening information will be listed. Rescreened patients will keep the same patient number, as for the initial screening.

Unscheduled measurements will not be included in by-visit summaries but will contribute to the EOS value, or best/ worst case value where required (e.g. shift table).

Early termination data will be mapped to the next available visit number for by-visit summaries, as described in Section 6.4 of the SAP.

Post-randomization if ECG result is Abnormal, Clinically Significant, then triplicate ECGs should be provided.

Listings will include scheduled, unscheduled, retest and early discontinuation data.

#### **6.4.** WINDOWING CONVENTIONS

Each visit (except for Day 1 visit) will have a±10 days window. No visit windowing will be applied during the analysis to the data that is only collected at scheduled site visits for patients that have completed the study, and therefore the data will be presented as per the visit reported in the database.

For endpoints based on 12 hour spirometry data, (FEV1 AUC0-12h, FEV1 evening trough and FEV1AUC6-12h), data collected at visits with 12 hour spirometries will be included in the analysis regardless of the timepoint it was generated. Hence, no windowing convention applied to these endpoints.

For the patients that discontinued from the study, the End of Study (EOS) visit will be windowed to the corresponding visit, based on the study day, for questionnaire, spirometry and rescue medication data. The EOS visit can only be windowed to a visit that is missing or has a missing result. The rules for the windowing are described below.





Statistical Analysis Plan


- For spirometry raw data and derived data that happens at every visit, windowing will be done
  as per the corresponding visits.
  - Day 1 = Day 1
  - Week 6 = after Day 1 and up to and including Day 53
  - Week 12 = after Day 53 and up to and including Day 95
  - Week 24= after Day 95 and up to and including Day 179
- For spirometry derived data that only happen at certain visits, windowing will be done for the corresponding visits.
  - For morning trough:
    - Week 6 = after Day 1 and up to and including Day 53
    - Week 12 = after Day 53 and up to and including Day 95
    - Week 24= after Day 95 and up to and including Day 179

•

- For rescue medication data, E-RS/EXACT-PRO, e-diary data and COPD exacerbation, windowing will be done as per the corresponding visits. Specifically, rescue medication data, E-RS/EXACT-PRO, e-diary data windowing conventions will be up to Week 24 whilst COPD exacerbation will be up to Week 48.
  - For patients who completed the study or who discontinue study medication but continue in the study:
- · Week 24 subset:
  - Week 1 = Actual study Day of Week 24 visit minus 168 days (inclusive) up to and including actual study day of week 24 visit minus 161 days
  - Week 2 = Actual study Day of Week 24 visit minus 161 days up to and including actual study day of week 24 visit minus 154 days
  - Week 3 = Actual study Day of Week 24 visit minus 154 days up to and including actual study day of week 24 visit minus 147 days
  - Week 4 = Actual study Day of Week 24 visit minus 147 days up to and including actual study day of week 24 visit minus 140 days
  - Week 5 = Actual study Day of Week 24 visit minus 140 days up to and including actual study day of week 24 visit minus 133 days
  - Week 6 = Actual study Day of Week 24 visit minus 133 days up to and including actual study day of week 24 visit minus 126 days
  - Week 7 = Actual study Day of Week 24 visit minus 126 days up to and including actual study day of week 24 visit minus 119 days
  - Week 8 = Actual study Day of Week 24 visit minus 119 days up to and including actual study day of week 24 visit minus 112 days
  - Week 9 = Actual study Day of Week 24 visit minus 112 days up to and





Statistical Analysis Plan


- including actual study day of week 24 visit minus 105 days
- Week 10 = Actual study Day of Week 24 visit minus 105 days up to and including actual study day of week 24 visit minus 98 days
- Week 11 = Actual study Day of Week 24 visit minus 98 days up to and including actual study day of week 24 visit minus 91 days
- Week 12 = Actual study Day of Week 24 visit minus 91 days up to and including actual study day of week 24 visit minus 84 days
- Week 13 = Actual study Day of Week 24 visit minus 84 days up to and including actual study day of week 24 visit minus 77 days
- Week 14 = Actual study Day of Week 24 visit minus 77 days up to and including actual study day of week 24 visit minus 70 days
- Week 15 = Actual study Day of Week 24 visit minus 70 days up to and including actual study day of week 24 visit minus 63 days
- Week 16 = Actual study Day of Week 24 visit minus 63 days up to and including actual study day of week 24 visit minus 56 days
- Week 17 = Actual study Day of Week 24 visit minus 56 days up to and including actual study day of week 24 visit minus 49 days
- Week 18 = Actual study Day of Week 24 visit minus 49 days up to and including actual study day of week 24 visit minus 42 days
- Week 19 = Actual study Day of Week 24 visit minus 42 days up to and including actual study day of week 24 visit minus 35 days
- Week 20 = Actual study Day of Week 24 visit minus 35 days up to and including actual study day of week 24 visit minus 28 days
- Week 21 = Actual study Day of Week 24 visit minus 28 days up to and including actual study day of week 24 visit minus 21 days
- Week 22 = Actual study Day of Week 24 visit minus 21 days up to and including actual study day of week 24 visit minus 14 days
- Week 23 = Actual study Day of Week 24 visit minus 14 days up to and including actual study day of week 24 visit minus 7 days
- Week 24 = Actual study Day of Week 24 visit minus 7 days up to and including actual study day of week 24 visit
- Week 48 subset:
- Week 1 = Actual study Day of Week 48 visit minus 336 days (inclusive) up to and including actual study day of week 48 visit minus 329 days
- Week 2 = Actual study Day of Week 48 visit minus 329 days up to and including actual study day of week 48 visit minus 322 days
- Week 3 = Actual study Day of Week 48 visit minus 322 days up to and including actual study day of week 48 visit minus 315 days



Statistical Analysis Plan


- Week 4 = Actual study Day of Week 48 visit minus 315 days up to and including actual study day of week 48 visit minus 308 days
- Week 5 = Actual study Day of Week 48 visit minus 308 days up to and including actual study day of week 48 visit minus 301 days
- Week 6 = Actual study Day of Week 48 visit minus 301 days up to and including actual study day of week 48 visit minus 294 days
- Week 7 = Actual study Day of Week 48 visit minus 294 days up to and including actual study day of week 48 visit minus 287 days
- Week 8 = Actual study Day of Week 48 visit minus 287 days up to and including actual study day of week 48 visit minus 280 days
- Week 9 = Actual study Day of Week 48 visit minus 280 days up to and including actual study day of week 48 visit minus 273 days
- Week 10 = Actual study Day of Week 48 visit minus 273 days up to and including actual study day of week 48 visit minus 266 days
- Week 11 = Actual study Day of Week 48 visit minus 266 days up to and including actual study day of week 48 visit minus 259 days
- Week 12 = Actual study Day of Week 48 visit minus 259 days up to and including actual study day of week 48 visit minus 252 days
- Week 13 = Actual study Day of Week 48 visit minus 252 days up to and including actual study day of week 48 visit minus 245 days
- Week 14 = Actual study Day of Week 48 visit minus 245 days up to and including actual study day of week 48 visit minus 238 days
- Week 15 = Actual study Day of Week 48 visit minus 238 days up to and including actual study day of week 48 visit minus 231 days
- Week 16 = Actual study Day of Week 48 visit minus 231 days up to and including actual study day of week 48 visit minus 224 days
- Week 17 = Actual study Day of Week 48 visit minus 224 days up to and including actual study day of week 48 visit minus 217 days
- Week 18 = Actual study Day of Week 48 visit minus 217 days up to and including actual study day of week 48 visit minus 210 days
- Week 19 = Actual study Day of Week 48 visit minus 210 days up to and including actual study day of week 48 visit minus 203 days
- Week 20 = Actual study Day of Week 48 visit minus 203 days up to and including actual study day of week 48 visit minus 196 days
- Week 21 = Actual study Day of Week 48 visit minus 196 days up to and including actual study day of week 48 visit minus 189 days
- Week 22 = Actual study Day of Week 48 visit minus 189 days up to and including actual study day of week 48 visit minus 182 days
- Week 23 = Actual study Day of Week 48 visit minus 182 days up to and





Statistical Analysis Plan 

- including actual study day of week 48 visit minus 175 days
- Week 24 = Actual study Day of Week 48 visit minus 175 days up to and including actual study day of week 48 visit minus 168 days
- Week 25 = Actual study Day of Week 48 visit minus 168 days up to and including actual study day of week 48 visit minus 161 days
- Week 26 = Actual study Day of Week 48 visit minus 161 days up to and including actual study day of week 48 visit minus 154 days
- Week 27 = Actual study Day of Week 48 visit minus 154 days up to and including actual study day of week 48 visit minus 147 days
- Week 28 = Actual study Day of Week 48 visit minus 147 days up to and including actual study day of week 48 visit minus 140 days
- Week 29 = Actual study Day of Week 48 visit minus 140 days up to and including actual study day of week 48 visit minus 133 days
- Week 30 = Actual study Day of Week 48 visit minus 133 days up to and including actual study day of week 48 visit minus 126 days
- Week 31 = Actual study Day of Week 48 visit minus 126 days up to and including actual study day of week 48 visit minus 119 days
- Week 32 = Actual study Day of Week 48 visit minus 119 days up to and including actual study day of week 48 visit minus 112 days
- Week 33 = Actual study Day of Week 48 visit minus 112 days up to and including actual study day of week 48 visit minus 105 days
- Week 34 = Actual study Day of Week 48 visit minus 105 days up to and including actual study day of week 48 visit minus 98 days
- Week 35 = Actual study Day of Week 48 visit minus 98 days up to and including actual study day of week 48 visit minus 91 days
- Week 36 = Actual study Day of Week 48 visit minus 91 days up to and including actual study day of week 48 visit minus 84 days
- Week 37 = Actual study Day of Week 48 visit minus 84 days up to and including actual study day of week 48 visit minus 77 days
- Week 38 = Actual study Day of Week 48 visit minus 77 days up to and including actual study day of week 48 visit minus 70 days
- Week 39 = Actual study Day of Week 48 visit minus 70 days up to and including actual study day of week 48 visit minus 63 days
- Week 40 = Actual study Day of Week 48 visit minus 63 days up to and including actual study day of week 48 visit minus 56 days
- Week 41 = Actual study Day of Week 48 visit minus 56 days up to and including actual study day of week 48 visit minus 49 days
- Week 42 = Actual study Day of Week 48 visit minus 49 days up to and including actual study day of week 48 visit minus 42 days



Statistical Analysis Plan


- Week 43 = Actual study Day of Week 48 visit minus 42 days up to and including actual study day of week 48 visit minus 35 days
- Week 44 = Actual study Day of Week 48 visit minus 35 days up to and including actual study day of week 48 visit minus 28 days
- Week 45 = Actual study Day of Week 48 visit minus 28 days up to and including actual study day of week 48 visit minus 21 days
- Week 46 = Actual study Day of Week 48 visit minus 21 days up to and including actual study day of week 48 visit minus 14 days
- Week 47 = Actual study Day of Week 48 visit minus 14 days up to and including actual study day of week 48 visit minus 7 days
- Week 48 = Actual study Day of Week 48 visit minus 7 days up to and including actual study day of week 48 visit
- For patients who discontinue the study before Week 24 (for 24-week stratum) or Week 48 (for 48-week stratum):
  - Week 24 subset:
  - Week 1 = on or after Day 1 and up to and including Day 8
  - Week 2 = after Day 8 and up to and including Day 15
  - Week 3 = after Day 15 and up to and including Day 22
  - Week 4 = after Day 22 and up to and including Day 29
  - Week 5 = after Day 29 and up to and including Day 36
  - Week 6 = after Day 36 and up to and including Day 43 Week 7 = after Day 43 and up to and including Day 50
  - Week 8 = after Day 50 and up to and including Day 57
  - Week 9 = after Day 57 and up to and including Day 64
  - Week 10 = after Day 64 and up to and including Day 71
  - Week 11 = after Day 71 and up to and including Day 78

  - Week 12 = after Day 78 and up to and including Day 85
  - Week 13 = after Day 85 and up to and including Day 92
  - Week 14 = after Day 92 and up to and including Day 99
  - Week 15 = after Day 99 and up to and including Day 106
  - Week 16 = after Day 106 and up to and including Day 113
  - Week 17 = after Day 113 and up to and including Day 120
  - Week 18 = after Day 120 and up to and including Day 127 Week 19 = after Day 127 and up to and including Day 134

  - Week 20 = after Day 134 and up to and including Day 141
  - Week 21 = after Day 141 and up to and including Day 148
  - Week 22 = after Day 148 and up to and including Day 155
  - Week 23 = after Day 155 and up to and including Day 162





Statistical Analysis Plan


- Week 24 = after Day 162 and up to and including Day 169
- •
- Week 48 subset:
- Week 1 = on or after Day 1 and up to and including Day 8
- Week 2 = after Day 8 and up to and including Day 15
- Week 3 = after Day 15 and up to and including Day 22
- Week 4 = after Day 22 and up to and including Day 29
- Week 5 = after Day 29 and up to and including Day 36
- Week 6 = after Day 36 and up to and including Day 43
- Week 7 = after Day 43 and up to and including Day 50
- Week 8 = after Day 50 and up to and including Day 57
- Week 9 = after Day 57 and up to and including Day 64
- Week 10 = after Day 64 and up to and including Day 71
- Week 11 = after Day 71 and up to and including Day 78
- Week 12 = after Day 78 and up to and including Day 85
- Week 13 = after Day 85 and up to and including Day 92
- Week 14 = after Day 92 and up to and including Day 99
- Week 15 = after Day 99 and up to and including Day 106
- Week 16 = after Day 106 and up to and including Day 113
- Week 17 = after Day 113 and up to and including Day 120
- Week 18 = after Day 120 and up to and including Day 127
- Week 19 = after Day 127 and up to and including Day 134
- Week 20 = after Day 134 and up to and including Day 141
- Week 21 = after Day 141 and up to and including Day 148
- Week 22 = after Day 148 and up to and including Day 155
- Week 23 = after Day 155 and up to and including Day 162
- Week 24 = after Day 162 and up to and including Day 169
- Week 25 = after Day 169 and up to and including Day 176
- Week 26 = after Day 176 and up to and including Day 183
- Week 27 = after Day 183 and up to and including Day 190
- Week 28 = after Day 190 and up to and including Day 197
- Week 29 = after Day 197 and up to and including Day 204
- Week 30 = after Day 204 and up to and including Day 211
- Week 31 = after Day 211 and up to and including Day 218
- Week 32 = after Day 218 and up to and including Day 225
- Week 33 = after Day 225 and up to and including Day 232
- Week 34 = after Day 232 and up to and including Day 239
- Week 35 = after Day 239 and up to and including Day 246
- Week 36 = after Day 246 and up to and including Day 253



Statistical Analysis Plan


- Week 37 = after Day 253 and up to and including Day 260
- Week 38 = after Day 260 and up to and including Day 267
- Week 39 = after Day 267 and up to and including Day 274
- Week 40 = after Day 274 and up to and including Day 281
- Week 41 = after Day 281 and up to and including Day 288
- Week 42 = after Day 288 and up to and including Day 295
- Week 43 = after Day 295 and up to and including Day 302
- Week 44 = after Day 302 and up to and including Day 309
- Week 45 = after Day 309 and up to and including Day 316
- Week 46 = after Day 316 and up to and including Day 323
- Week 47 = after Day 323 and up to and including Day 330
- Week 48 = after Day 330 and up to and including Day 337

## 6.5. STATISTICAL TESTS

In general, unless stated otherwise, continuous variables will be summarized using descriptive statistics (number of patients, mean, standard deviation [SD], median, minimum and maximum values) and for categorical (nominal) variables, the number and percentage of patients will be used.

The default significant level will be 5%; CIs will be 95% and all tests will be two-sided, unless otherwise specified in the description of the analyses.

#### 6.6. COMMON CALCULATIONS

- Change from baseline: Test Value at Visit X Baseline Value
- Percentage change from baseline:

Test Value at Visit X – Baseline Value

Baseline Value

\* 100%

## 6.7. ACTUAL TREATMENT

Once the study unblinds, the patient's actual treatment will be assigned based on the most frequent medication they have received throughout the study. Patients are only expected to receive either 3 mg of ensifentrine, or placebo. The external vendor, Cenduit, will provide the Material List document after confirmation of a DBL. This document will contain the kit numbers, which will be merged with the site data to obtain the treatment that was dispensed at each visit.

If a patient takes more than one medication and the ratio of actual treatments taking the placebo



Statistical Analysis Plan


and ensifentrine is the same, then the patient will be assigned ensifentrine.

#### 6.8. SOFTWARE VERSION

All analyses will be conducted using SAS version 9.4 or higher.

#### 6.9. STRATA CALCULATIONS

There are three separate stratification factors used: treatment duration (48 or 24 weeks), background maintenance therapy strata and smoking strata. For all factors planned and actual will be created.

For treatment duration strata:

- Planned As recorded in the Cenduit report.
- Actual The actual treatment duration in which the patient consented to in the Patient Consent form
- In case when the randomized treatment duration stratum does not match with the treatment duration the patient consented to, the patient will be assigned to the stratum they consented to.

For background maintenance therapy strata:

- Planned As recorded in the Cenduit report.
- Actual As recorded in the "Concomitant medications" eCRF page: Patients that take
  LAMA or LABA (or LAMA/ICS or LABA/ICS) medication with start date being before or
  on randomization date and end date is either ongoing/post-randomization are classified as
  being on background maintenance therapy strata. Patients that do not meet this criteria will
  be classified as "No".

## For smoking strata:

- Planned As recorded in the Cenduit report.
- Actual As recorded in the "COPD and Smoking History" eCRF page.

#### 6.10. Russian Laboratories

At the start of the study, the laboratory data collected from Russian sites were to be collected from the central sources. However, from 23 March 2022, which is the date of the first collection





Statistical Analysis Plan


from local laboratory reported in Inform, the data have been coming from either central or local sources. These sources use different ranges for laboratory parameters.

The laboratory ranges will be entered by the sites directly into the eCRF if done by a local laboratory or if received by a data transfer from InVitro laboratories. All units will be converted to conventional or SI units for consistency of the original Q2 laboratory tests received prior to the implementation of using InVitro or the local laboratories to indicate low/normal/high categories. Any alert or flag variable in the received data that indicates its category will not be used.

## 7. STATISTICAL CONSIDERATIONS

# 7.1. ADJUSTMENTS FOR COVARIATES AND FACTORS TO BE INCLUDED IN ANALYSES

The following covariates and factors are used in the analyses. For details of their inclusion in the models, see the specific analysis section.

Fixed effects: treatment (ensifentrine, placebo), region (Asia, Europe, North America), visit (Day 1, Week 6, Week 12, Week 18, Week 24), visit\*treatment, stable background maintenance of LABA or LAMA (or LAMA/ICS or LABA/ICS) therapy use (yes, no), cigarette smoking (current, former)

Random effect: patient Covariate: baseline

In case when the analysis model does not converge, the factor that causes it will be removed from the model.

## 7.2. MULTICENTER STUDIES

This study will be conducted by multiple investigators at multiple centers internationally. Randomization to treatment arms is not stratified by country/ center.

When specified, statistical analysis will be adjusted for geographic region. Geographic region will be categorized as shown in Table 3.





Statistical Analysis Plan


Table 3: Geographic Regions

| Geographic Region | Country |
|---|---|
| Asia | Republic of Korea |
| Europe | Bulgaria, Czech Republic, Germany, Greece, Hungary, Poland,<br>Romania, Russian Federation, Slovakia, United Kingdom |
| North America | United States |

## 7.3. MISSING DATA

Missing safety data will not be imputed.

All data collected during the scheduled visits for patients on-treatment and off-treatment, for patients with treatment withdrawal, as well as the end-of-study visits for patients withdrawing from the study will be used for analysis performed on the mITT and that the remaining missing values will be handled as described in Sections 16.1.2, 16.2.2 and 16.3.2 of the SAP.

#### 7.4. MULTIPLE COMPARISONS/ MULTIPLICITY

To address multiplicity in the analysis of the endpoints, statistical testing of the primary endpoint and key secondary endpoints will be done in the hierarchical order (listed below). Initially the primary endpoint will be checked to see if comparison between active treatment and placebo is statistically significant. If yes, the first key secondary endpoint will be evaluated. If yes, the next key secondary endpoint will be evaluated. This process will continue until either all endpoints are evaluated, or if one of the endpoints' comparison is not significant.

Order of the endpoints that will be used for the hierarchical testing:

- 1. Change from baseline FEV<sub>1</sub> to FEV<sub>1</sub> AUC<sub>0-12h</sub> at Week 12
- Change from baseline FEV<sub>1</sub> to peak FEV<sub>1</sub> at Week 12
- 3. Change from baseline (i.e. mean over the last 7 days of run-in) to the mean weekly value at Week 24 in COPD symptoms, as measured by daily diary (E-RS<sup>TM</sup>:COPD)
- 4. Change from baseline in the SGRQ total score at Week 24
- 5. Change from baseline FEV1 to morning trough FEV1 at Week 12
- 6. Change from baseline FEV1 to average FEV1 AUC0-4h at Week 12
- 7. Proportion of SGRQ responders at Week 24

## 7.5. EXAMINATION OF SUBGROUPS

Subgroup analyses will be conducted as stated in the efficacy analysis and disposition sections.



Statistical Analysis Plan


Primary aim for the subgroup analysis is to check whether there are differences in treatment effect between strata or subgroups, which will be tested through interaction. For each analysis by subgroup the results will be summarized as follows:

- Complete data with added fixed effect to the model: subgroup\*treatment.
- Data split by subgroup using the main model.

The following subgroups will be assessed and described within the analysis Sections 16.1.4 and 16.2.4 of the SAP.

- Gender at birth:
  - o Female
  - Male
- Age-class (years):
  - 0 <65
  - o ≥65
- Region
  - Asia
  - Europe
  - North America
- Actual Background medication strata
  - o Yes
  - o No
- Actual Smoking strata
  - o Current
  - o Former
- Actual ICS use
  - o Yes
  - o No
- · Known chronic bronchitis
  - o Yes
  - o No
- FEV<sub>1</sub> reversibility at screening ( $\geq$ 12% and  $\geq$ 200mL increase in FEV<sub>1</sub>)
  - o Yes
  - o No
- COPD severity





Statistical Analysis Plan


- o Mild (post-bronchodilator dose  $FEV_1 \ge 80\%$  predicted)
- Moderate ( $50\% \le baseline FEV_1 < 80\% predicted$ )
- Severe (30%  $\leq$  baseline FEV<sub>1</sub>  $\leq$ 50% predicted)
- Very severe (baseline FEV<sub>1</sub> <30% predicted)</li>

All the four categories of COPD severity will be included in the patient disposition presentations. However, when used in efficacy analysis, only the two subgroups with moderate and severe patients will be used in the analysis models.

## 8. OUTPUT PRESENTATIONS

Appendix 1 shows conventions for presentation of data in outputs.

The shells document provided with this SAP describe the presentations for this study and therefore the format and content of the summary tables, figures, and listings to be provided by IQVIA Biostatistics.

## 9. DISPOSITION AND WITHDRAWALS

All patients who provide informed consent will be accounted for in this study. Cenduit will be the primary source for the randomization information.

## 9.1. DISPOSITION

Patient disposition and withdrawals will be presented for the RND set using frequency counts and percentages by treatment. Patients who withdrew after week 24 (for 24-week stratum) and after week 48 (for 48-week stratum) will be included in the tables. Separate tables will be provided for patient disposition by treatment and by visit. The following patient sets will be presented per stratum and overall:

- · Number of patients rescreened with approval
- · Number of patients rescreened without approval
- · Number of patients randomized
- · Number of patients randomized and treated
- Number of patients who completed the full study, including follow-up visit
- Number of patients who completed treatment period in the study, up to Week 24 (overall, 24-week stratum and 48-week stratum)
- Number of patients who completed treatment period on study medication (overall, 24-





Statistical Analysis Plan


- week stratum and 48-week stratum)
- Number of patients who discontinued the study medication (overall, 24-week stratum and 48-week stratum)
- Primary reason for early study medication discontinuation
- Number of patients who withdrew from the study (overall, 24-week stratum and 48-week stratum)
- Primary reason for early study withdrawal

Study medication and study discontinuation/completion of patients will be presented by the date of the "End of Treatment/Disposition" page of the eCRF. The date of study discontinuation/completion will be last available date within eCRF and the date of study medication completion will be identified from End of Treatment page of the eCRF.

The number of study discontinuation and study medication discontinuation before 24 weeks visit (all subjects) and before 48 weeks (48-week stratum only) will be summarized by treatment group and analyzed and presented through Kaplan-Meier plot using log-rank test, as described in Section **** of the SAP.

Time to study medication discontinuation by subgroups of actual background medication strata and actual smoking strata will be presented through Kaplan-Meier plot.

Reasons for exclusion from each analysis set, as well as patients not meeting eligibility and randomization criteria will be presented for the ENR set with patients classified according to the randomized treatment. Patients not randomized will be presented in a separate category.

#### 9.1.1. DERIVATIONS

Study day of early study medication discontinuation = Last day of study medication intake - First day of study medication intake + 1.

Study day of early study discontinuation = Last day in the study - First day of study medication intake + 1.

Visit for discontinuation will be presented using six subgroups (Not treated,  $\geq$  day 1 and  $\leq$  week 6, > week 6 and  $\leq$  week 12, > week 12 and  $\leq$  week 24, > week 24 and  $\leq$  week 36, > week 36 and  $\leq$  week 48), using the corresponding visit day windowing:

week 6 = study day 53


Statistical Analysis Plan


- week 12 = study day 95
- week 24 = study day 179
- week 36 = study day 263
- week 48 = study day 336

## 9.2. PROTOCOL DEVIATIONS

PDs will be defined in the BDR report and the list will be finalized before the DBL. Identified PDs that affect the BDR and analysis populations will be finalized before DBL.

## 9.3. EVALUATION INCLUDING EXCLUDED SITES

Sites were removed from the Randomized set. As a check of this exclusion, the patient disposition will be performed in the Extended Randomized set.

## 10. DEMOGRAPHIC AND OTHER BASELINE CHARACTERISTICS

Demographic data and other baseline characteristics will be presented for the RND. If there is a difference in patients between RND and mITT population, then demographic data and other baseline characteristics will also be presented for mITT.

Demographic data and other baseline characteristics will also be presented by subgroups of actual background medication strata and actual smoking strata for mITT.

No statistical testing is planned be carried out for demographic or other baseline characteristics. The following demographic and other baseline characteristics will be reported for this study:

- Age (years)
- Age-class (years) (<65, ≥65)</li>
- · Gender at birth
- Ethnicity (Hispanic or Latino, Not Hispanic or Latino (subgroup for rest of categories), Not Reported)
- Race
- Country
- Weight (kg)
- Height (cm)
- BMI (kg/m<sup>2</sup>)



Statistical Analysis Plan


- FEV<sub>1</sub> reversibility at screening (yes, no)
- Modified Medical Research Council (mMRC) questionnaire score
- Pre- and post-bronchodilator FEV<sub>1</sub> (both in liters and in percentage of predicted normal)
- Post-bronchodilator FEV<sub>1</sub>/forced vital capacity (FVC)
- Time since initial diagnosis of COPD (years)
- Background medication strata [yes (subgroup for yes: LAMA, LAMA/ICS, LABA, LABA/ICS), no] –actual
- Known to have Chronic Bronchitis (yes, no)
- Known to have Emphysema (yes, no)
- Smoking strata (current, former) –actual recorded in the eCRF
- · Number of cigarettes per day, Number of years smoking, Number of Pack Years
- COPD severity based on post-bronchodilator FEV1 (Mild, Moderate, Severe, Very severe)

## 10.1. DERIVATIONS

- BMI (kg/ $m^2$ ) = weight (kg)/height (m)<sup>2</sup>
- Time since initial diagnosis of COPD = (date of consent date first diagnosed)/365.25
- Pack Years = Number of packs per day x number of years smoking

Reversibility status is calculated based on pre-bronchodilator and post-bronchodilator FEV<sub>1</sub> values taken at Screening. If patient has increase of  $\geq$ 12% and  $\geq$ 200mL then patient is reversible, else patient is non-reversible.

Age (years) collected in the eCRF will be used for the analysis.

Pack Years is automatically calculated in the eCRF and this value will be used in the summaries. COPD severity will be derived as follows based on post-bronchodilator screening spirometry:

- Mild: post-bronchodilator FEV<sub>1</sub> ≥ 80% predicted
- Moderate: 50% ≤ post-bronchodilator FEV<sub>1</sub> < 80% predicted</li>
- Severe: 30% ≤ post-bronchodilator FEV<sub>1</sub> <50% predicted</li>
- Very severe: post-bronchodilator FEV<sub>1</sub> <30% predicted</li>

10.2. EVALUATION INCLUDING EXCLUDED SITES

As a check of the exclusion of sites from the mITT, the demography and baseline disease characteristics will be performed in the mITT Extended.

Copyright © 2009, 2010, 2012, 2016, 2018, 2019 IQVIA. All rights reserved. The contents of this document are confidential and proprietary to IQVIA Holdings Inc. and its subsidiaries. Unauthorized use, disclosure or reproduction is strictly prohibited.

Statistical Analysis Plan


## 11. SURGICAL AND MEDICAL HISTORY

Surgical and Medical History information will be presented for the SAF set.

- Surgical History will be coded using the Medical Dictionary for Regulatory Activities
  (MedDRA) central coding dictionary. The version of MedDRA to be used will be specified
  prior to database lock. Data captured on the "Surgical Procedure History" page of the eCRF
  will be presented by System Organ Class (SOC) and Preferred Term (PT) for each treatment
  group.
- Medical History will be coded using MedDRA central coding dictionary. The version of MedDRA to be used will be specified prior to database lock.
  - Medical History conditions, captured on the "Medical History" page of the eCRF, are defined as those conditions which stop prior to or at Screening visit and will be presented by SOC and PT for each treatment group.

## 12. CONCOMITANT ILLNESSES

Concomitant Illnesses will be presented for the SAF set.

- Concomitant Illnesses will be coded using MedDRA central coding dictionary. The version
  of MedDRA to be used will be specified prior to database lock.
  - Concomitant Illnesses, captured on the "Medical History" page of the eCRF, are conditions which started prior to the first treatment dose and are ongoing at the date of first treatment dose, and will be presented by SOC and PT for each treatment group.

## 13. MEDICATIONS

Prior, prior concomitant and concomitant medications will be presented separately for the SAF set and coded using the World Health Organization (WHO) drug code and summarized by Anatomical Therapeutic Clinical Classification System (ATC) levels 1, 2 and 4.

Possible therapeutic subgroups include ICS, LABA, LAMA, corticosteroids, short-acting B2 agonist, short-acting anti-muscarinic and combinations specified below, which are defined in a separate spreadsheet provided by the medical data reviewer. Combinations to be analyzed:

- 1. Oral or intravenous (IV) Corticosteroids
- 2. Oral or IV Corticosteroid & Other combinations
- 3. LAMA
- 4. LAMA/LABA



Statistical Analysis Plan


- LAMA & OTHER COMBINATIONS
- 6. LABA
- 7. LABA & Other combinations
- 8. ICS/LAMA/LABA or ICS/LABA/LAMA
- 9. ICS/LAMA
- 10. ICS/LABA
- 11. ICS & Other Combinations
- 12. SABA/Short-Acting Anti-Muscarinic
- 13. SABA
- 14. SABA & other combinations
- 15. SABA/ICS
- 16. SABA/ Corticosteroid
- 17. Short-Acting Anti-Muscarinic

See Appendix 2 for handling of partial dates for medications, in the case where it is not possible to define a medication as prior, concomitant, or post treatment, the medication will be classified by the worst case; i.e. concomitant.

- 'Prior' medications are medications which started prior to the first dose of study medication and stopped prior to the first dose of study medication.
- 'Prior Concomitant' medications are medications which started prior to the first dose of study
  medication and ended on or after the date of first dose of study medication or were ongoing
  at the end of the study.
- 'Concomitant' medications are medications which:
  - started on or after the first dose of study medication and started no later than last day of study medication intake,
  - AND ended on or after the date of first dose of study medication or were ongoing at the end of the study.
- 'Post' medications are medications which started from the day after the last dose of study medication.

Prior, prior concomitant and concomitant COPD medications will be presented separately for the SAF set. COPD medications are those provided by medical review and will be presented as preferred term and ATC levels 1, 2 and 4.

Data captured on the "Concomitant Medications" page of the eCRF will be presented for each treatment group. Patients with multiple medications within an ATC/ therapeutic subgroup will only be counted once for that level.





Statistical Analysis Plan


Oxygen therapy and CPAP will be listed separately to other medications. Oxygen therapy is defined by ATC code: "V03AN" and route is not Oral; CPAP is defined by ATC code: "R07AX" and route is not Oral.

## 14. STUDY MEDICATION EXPOSURE

Exposure to study medication in days will be presented for the SAF set.

The dates of first dose of study medication administration will be taken from the "Drug Exposure" page of the eCRF (Day 1). The date of last dose of study medication administration will be taken as the latest date among all from the "Drug Exposure" and "Drug Exposure – Evening Blinded Study Medication Clinic Dosing" pages of the eCRF. If no drug exposure were made at last visit and the dispensed drug supply was insufficient to cover use up to last visit, the last exposure day will be set to the day the drug supply should have been empty if patient had been compliant to twice daily regimen. Interruptions and compliance are not taken into account for duration of exposure.

Study medication exposure will be presented using summary statistics by total number of days, and using frequency counts by subgroups: 1-42 days, 43-84 days, 85-126 days, 127-168 days, 169-210 days, 211-252 days, 253-294 days, 295-336 days, and >336 days.

#### 14.1. DERIVATIONS

Duration of exposure (days) = date of last study medication administration – date of first study medication administration + 1.

## 15. COMPLIANCE

Compliance to study medication based on dispensed and returned unused ampules and secondarily based on e-Diary entries will be presented for the SAF set.

Compliance will be presented for 24-week and 48-week strata separately using summary statistics by time intervals (Day 1 to Week 12, Weeks 12-24, Weeks 24-48, and full study length), as well as using frequency counts by subgroups: <50%, 50-70%, 70-80%, 80-90%, 90-100% and >100%.

## 15.1. STUDY MEDICATION COMPLIANCE

Study medication compliance will be summarized by treatment group in 2 ways:

The number of ampules dispensed and unused returned will be taken from "Drug



Copyright © 2009, 2010, 2012, 2016, 2018, 2019 IQVIA. All rights reserved. The contents of this document are confidential and proprietary to IQVIA Holdings Inc. and its subsidiaries. Unauthorized use, disclosure or reproduction is strictly prohibited.



Statistical Analysis Plan


Accountability" page of the eCRF.

· Drug intake as recorded in the e-diary.

Patient is non-compliant, for study medication intake collected through the number of ampules dispensed/returned, if identified as taking less than or equal to 70% of blinded study medication during the period Day 1 to Week 12, or less than or equal to 50% over the study (Day 1 to Week 24 for the 24-week stratum, Day 1 to Week 48 for the 48-week stratum). Calculations will not include time after treatment withdrawal.

#### 15.1.1. DERIVATIONS

Compliance with study medication will be calculated on the number of ampules count (total dispensed – total returned) divided by the prescribed number of ampules expressed as a percentage, see calculations below.

Patient should take the study medication twice daily and record it in their e-Diary apart from Week 24 visit when patient's last dose will be in the morning.

Patients are dispensed ampules at Visit X and return at Visit Y, however in the eCRF returned ampules will be recorded under Visit X.

• For time interval compliance to study medication will be calculated as follows:

([N of Ampules dispensed at Visit X] – [N of Ampules returned at Visit Y])

Denominator1 \* 100

Where Denominator1 is calculated with the following rules:

- $\circ$  N<sub>1</sub> = Number of ampules expected calculated based on total N of Ampules dispensed, taking into account 2 ampules per day, apart from last dose date for completed patients where we would only consider 1 ampule per day.
- For non-Week 24 (for the 24-week stratum) or non-Week 48 (for the 48-week stratum) (last week) return ampules visit: N<sub>2</sub> = Number of ampules between dispensing and returning visit calculated: {[Date of Visit Y] [Date of Dispensing at Visit X]+1}\* 2.
- For Week 24 (for the 24-week stratum) or Week 48 (for the 48-week stratum) (last week) return ampules visit: N<sub>2</sub> = Number of ampules between dispensing and returning visit calculated: {{[Date of Visit Y] [Date of Dispensing at Visit X]+1}\* 2}-1.
- o If  $N_1 \ge N_2$  then Denominator  $1 = N_2$ .
- o If  $N_1 < N_2$  then Denominator  $1 = N_1$ .





Statistical Analysis Plan


0

• Overall Compliance to study medication will be calculated as follows:

Where Denominator2 is calculated with the following rules:

- N<sub>1</sub> = Number of days calculated based on total N of Ampules dispensed, taking into account 2 ampules per day, apart from last dose date for completed patients where we would only consider 1 ampule per day.
- N<sub>2</sub> = Number of days between dispensing and returning visit calculated: {{[Date of Visit X(n)] [Date of Dispensing at Visit 1]+1}\* 2}-1.
- o If  $N_1 \ge N_2$  then Denominator  $2 = N_2$ .
- o If  $N_1 < N_2$  then Denominator  $2 = N_1$ .

For patients who permanently discontinue the study medication, the "Date of Visit X(n)"/ "Date of Visit Y" will be replaced by the last dose date of study medication, as specified in Section 14 of the SAP. Whereas for patients who completed study, the "Date of Visit X(n)"/ "Date of Visit Y" will be replaced by date of last dose.

Drug intake as recorded in the e-diary: percent of 'yes' responses. The denominator is the number of records for which the patient provided an answer (Yes or No) to drug intake questions (morning and evening) in the e-diary.

For time interval study medication e-diary compliance, use week's windowing conventions described in Section 6.4 of the SAP. For Week 24 (for the 24-week stratum), use study day assigned to determine the date for weeks required or the time intervals, Week 12 and Week 24. The compliance will be calculated as follows:

```
\frac{\left(\text{Week X}^* < \text{number of 'yes' responses entered in the eDiary} \leq \text{Week Y}\right)}{\left(\text{Week X}^* < \text{number of non} - \text{missing responses entered in the } e - \text{Diary} \leq \text{Week Y}\right)} * 100
```

\*If Week X = Day 1, update "<" to be "\le ". For the 24-week stratum, if Week Y is Week 24 and patient has completed treatment then the last entry we expect is in the morning. Patient should not log any entries from and including evening of Week 24.

Similarly for Week 48 visit for the 48-week stratum, determine the time intervals using study day as described above for Week 12, Week 24, and Week 48. As above, if Week Y is Week 48 and patient has completed treatment the last entry expected will be morning and no further log entry





Statistical Analysis Plan


should be done including the evening of Week 48.

#### 15.2. E-DIARY COMPLIANCE

The flow of the eDiary entries patient has to follow is:

- 1. E-RS
- 2. Study medication compliance
- 3. Background medication compliance (if applicable)
- 4. Rescue medication use

Based on this, we can assess if patient has been compliant with their E-RS questions, based on their study medication compliance and therefore no further E-RS compliance needs to be assessed.

#### 15.2.1. DERIVATIONS

E-diary compliance will be calculated as per the following. Use study day assigned to determine the date for each week, as per the windowing conventions described in Section 6.4 of the SAP:

$$\frac{\text{(Week X}^* < \text{number of days study medication data was entered in the } e - \text{Diary} \le \text{Week Y})}{\text{[Study Day at Week Y]} - \text{[Study Day at Week X}} * 100}$$

\*If Week X = Day 1, update "<" to be " $\leq$ ".



Statistical Analysis Plan


## 16. EFFICACY OUTCOMES

#### 16.1. PRIMARY EFFICACY

The primary efficacy analysis will be performed for the mITT population.

#### 16.1.1. PRIMARY EFFICACY VARIABLE & DERIVATION

The primary efficacy variable is change from baseline in  $FEV_1$  AUC<sub>0-12h</sub> at Week 12.  $FEV_1$  data captured in the eResearch Technology (ERT) database will be used for the model in determining baseline value and for AUC calculation.

#### 16.1.1.1. AUC<sub>0-T</sub>

Spirometry (FEV<sub>1</sub>) will be performed at Screening and the following time points during, each treatment:

- Day 1: ≤40 minutes pre-dose (2 measurements); 30 minutes, 1, 2 and 4 hours post-dose.
- Week 6 and Week 24: ≤40 minutes pre-dose; 30 minutes, 1, 2 and 4 hours post-dose.
- Week 12: ≤40 minutes pre-dose; 30 minutes, 1, 2, 4, 6, 8 and 12 hours post-dose.
- Early Termination and no Week 12 visit spirometry assessment: ≤40 minutes pre-dose; 30 minutes, 1, 2, 4, 6, 8 and 12 hours post-dose.
- Early Termination but with Week 12 visit spirometry assessment: ≤40 minutes pre-dose; 30 minutes, 1, 2 and 4 hours post-dose.

Baseline  $FEV_1$  is the mean of the two measurements taken before study medication on the day of first dosing, i.e.  $\leq$ 40 minutes pre-dose on Day 1.

The average effect will be calculated as the AUC divided by the length of the time interval of interest (for example, 12 hours for  $AUC_{0-12h}$  or 4 hours for  $AUC_{0-4h}$ ). AUC will be calculated using the trapezoidal method, as follows:

$$AUC = \frac{1}{2} \sum_{i=1}^{n-1} (T_{i+1} - T_i)(C_{i+1} + C_i)$$

Where Ti is the ith time value, Ci is the ith effect value, n is the number of time values. The change from the baseline  $FEV_1$  to average  $FEV_1$  (AUC) will be summarized and analyzed. If two last data points are missing the AUC is set to missing, that is for  $AUC_{0-12h}$  we require at least up to 8 hours of assessments and for  $AUC_{0-4h}$  we require at least up to 2 hours of assessments. This would mean if we only have 8 hours of assessments, then we would calculate  $AUC_{0-8h}$ , however it would still be labelled as  $AUC_{0-12h}$ . If there is no pre-dose measurement





Statistical Analysis Plan


available for the calculation of the AUC, then the AUC will not be calculated. The pre-dose measurement used in the calculation of AUC is the latest value measured  $\leq$ 40 minutes pre-dose. The pre-dose value will be used as time 0 when computing AUC<sub>0-T</sub>.

For AUC<sub>6-12h</sub> we require at least the 6-hour and 12-hour timepoint for analysis.

#### 16.1.2. MISSING DATA METHODS FOR PRIMARY EFFICACY VARIABLE

The main analysis for the primary endpoint will include estimates from missing data imputation described below. This is done to investigate the influence of missing data due to drop-outs. Only patients with non-missing baseline will be included in the analysis.

The primary analysis will be analyzed using MI based on the missing data assumption Missing at Random (MAR). This process will follow four steps:

- Partially impute the data for a monotone missing pattern with 100 as a number of imputations and "20905" as seed number. Employ the Markov Chain Monte Carlo (MCMC) method with treatment, region, background medication strata, smoking strata, baseline FEV<sub>1</sub> and average FEV<sub>1</sub> AUC<sub>0-12h</sub> at Week 12.
  - 1.1 The following SAS codes will be used:

```
proc mi data=<data1> out=<data2> nimpute=100 seed=20905;
   var <treatment> <region> <BackgroundMedStrata> <SmokingStrata>
   <baseline> <visits>;
   mcmc impute=monotone chain=multiple;
run;
```

2. Impute the monotone data using a regression imputation model. Apply by imputation using seed number "20905" with treatment, region, background medication strata, smoking strata, baseline FEV<sub>1</sub> and average FEV<sub>1</sub> AUC<sub>0-12h</sub> at Week 12.

#### The following SAS codes will be used:

- 3. Each multiple imputed dataset in Step 2 will be analyzed separately, as described in Section 16.1.3 of the SAP.
- 4. The estimates (LS means, SE, CI, and p-value) from the model analysis in Step 3 will be combined using Rubin's combination rules for statistical inference.





Statistical Analysis Plan


Sensitivity analysis will be done using:

- Average imputation will be based on data collected on treatment at required visit, or at early termination visit. This will be done on patient level. If there is no such data available, impute with average change from baseline for the particular visit in the opposite randomized treatment group.
- Tipping point approach will repeat the ANCOVA analysis, under Missing not at Random (MNAR) assumption, to assess the robustness of p-value significance. In case the original analysis will produce a p-value<0.05, then the imputed values will be adjusted by a value k (positive) added or subtracted (depending on what worsens the endpoint) to the endpoint of the patients in Ensifentrine group (worsening results) and added or subtracted (depending on what improves the endpoint) from the endpoint of the patients in placebo group (improving results). The value for k is determined by adjusting the bias starting with a value of 0.01 and increasing it with increments of 0.01 until p-value obtained from MI method is no longer statistically significant (p-value>0.05). Seed number used will be the same as for MI analysis, "20905". If the primary analysis is not significant (p-value>0.05), then the tipping point is reversed by determining value for k by adjusting the bias until p-value<0.05. If the p-value<0.05 with more improvement in the placebo group comparably to Ensifentrine group, then the tipping point is reversed by adjusting until there will be no more treatment difference between groups.

#### 16.1.3. PRIMARY ANALYSIS OF PRIMARY EFFICACY VARIABLE

The primary objective of this study is to test the hypothesis that there is a difference between ensifentrine in comparison with placebo.

The change from baseline FEV<sub>1</sub> to average FEV<sub>1</sub> AUC<sub>0-12h</sub> will be compared between ensifentrine and placebo using ANCOVA with fixed effects for treatment, region, background medication strata and smoking strata and baseline FEV<sub>1</sub> as covariate. Missing data will be imputed using imputation described in Section 16.1.2 of the SAP. The estimated treatment difference will be presented with 95% CI and associated p-value. Furthermore, SD will be presented for the treatment difference to check the sample size with 90% power. Summary statistics will be performed on the imputed values.

Model assumptions will be tested as per the following rules on the blinded data, before the DBL.

- Residual vs Predicted plots will be created to check residuals are uncorrelated and normally distributed.
- 2. Normality of the data will be checked using Kolmogorov-Smirnov normality test.





Statistical Analysis Plan


If any of the checks specified above fail the test, then alternative approaches will be discussed, including different ways of transposing data. The SAP will be updated to reflect any changes prior to DBL.

Only spirometry measurements with best test review (BTR) grades "Acceptable" and "Borderline Acceptable" are used in the analysis and baseline calculations.

#### 16.1.4. SENSITIVITY ANALYSIS OF PRIMARY EFFICACY VARIABLE

The primary endpoint will be presented for the following:

- Subgroup analysis will be performed by subgroups, including data imputation described in Sections 7.5 and 16.1.2 of the SAP, respectively.
- Observed data analysis will be performed by the following subgroups:
  - Analysis with no data imputation, including all patients with data collected, on treatment or not, and at required timepoint or at EOS visit (excluding patients with missing data).
  - Analysis with no data imputation, including only patients with data collected at the required visit while still on randomized treatment at scheduled visit, or at end of study visit within the visit window.
- Average imputation, as described in Section 16.1.2 of the SAP.
- Analysis with tipping point approach, as described in Section 16.1.2 of the SAP.
- Analysis with multiple imputation, as described in Sections 16.1.2 and 16.1.3 of the SAP, based on PP population.



Statistical Analysis Plan


#### 16.2. SECONDARY EFFICACY

The secondary efficacy analyses will be performed for the mITT population. These include:

- Change from baseline FEV<sub>1</sub> to peak FEV<sub>1</sub> on Day 1 and at Weeks 6, 12 and 24
- Change from baseline (i.e. mean over the last 7 days of run-in) to the mean weekly value at Weeks 6, 12 and 24 in COPD symptoms, as measured by daily diary (E-RS<sup>TM</sup>:COPD)
- Change from baseline in the SGRQ total score at Weeks 6, 12 and 24
- Change from baseline FEV<sub>1</sub> to morning trough FEV<sub>1</sub> at Weeks 6, 12 and 24
- Change from baseline FEV<sub>1</sub> to average FEV<sub>1</sub> AUC<sub>0-4h</sub> on Day 1 and at Weeks 6, 12 and 24
- Proportion of SGRQ responders at Weeks 6, 12 and 24
- Change from baseline (i.e. mean over the last 7 days of run-in) to the mean weekly value in the number of puffs of rescue medication at Weeks 6, 12 and 24
- TDI questionnaire at Weeks 6, 12 and 24
- Change from baseline FEV<sub>1</sub> to evening trough FEV<sub>1</sub> at Week 12

#### 16.2.1. SECONDARY EFFICACY VARIABLES & DERIVATIONS

#### 16.2.1.1. **Spirometry**

Spirometry measurement's best test time which is used in the analysis is measured in ERT and first time for spirometry measurements is measured in the eCRF and will be listed alongside the ERT best time.

Peak FEV<sub>1</sub> will be computed as the maximum value in the 4 hours after dosing (4 timepoints after dosing: 30 minutes, 1 hour, 2 hours and 4 hours). Baseline FEV<sub>1</sub> is the average of the two measurements taken before study medication on the day of first dosing, i.e.  $\leq$ 40 minutes pre-dose on Day 1.

Average FEV<sub>1</sub> AUC<sub>0-4h</sub> is calculated as described in Section 16.1.1.1 of the SAP.

Morning trough  $FEV_1$  is the last value collected prior to the morning dose.

Evening trough  $FEV_1$  is the value collected at the 12 hours post-morning dose timepoint and prior to the evening dose.

All measurements, including unscheduled measurements, within specified time period will be used for deriving parameters; for scheduled 12 hours post-morning dose measurement use regardless of being within specified time period.



Statistical Analysis Plan


#### 16.2.1.2. Questionnaires

## 16.2.1.2.1. E-RS<sup>TM</sup>:COPD

EXACT-Respiratory Symptoms for COPD (E-RS<sup>TM</sup>: COPD) data will be collected within EXACT-PRO questionnaire (consisting of 14 questions), as shown in Appendix 3. Please note that items 3, 8, 9, 10, 11 and 14 have separate scoring instructions, namely with the same raw score being assigned to several answer options. E-RS<sup>TM</sup>: COPD consists of 11 questions, with subdomains of: Breathlessness, Cough and Sputum, and Chest Symptoms. This data will be collected everyday throughout the duration of the study.

#### Calculating the score

E-RS subdomains:

- Breathlessness items 7, 8, 9, 10 and 11 (score range: 0-17)
- Cough and Sputum items 2, 3 and 4 (score range: 0-11)
- Chest Symptoms items 1, 5 and 6 (score range: 0-12)

The E-RS Total score is derived as the sum of the raw scores of the 11 items (score range: 0-40). Total and subdomain scores are derived weekly as the mean over the days within each window, as specified in the Section 6.4 of the SAP, using only days where data was recorded. Baseline is the mean over the 7 days prior to the first intake of study treatment, using only days where data was recorded. If less than 4 days of data are available for the week, the weekly mean is set to missing. Furthermore, all questions need to be answered to be evaluable for that day.

If a patient discontinued then use treatment study end date, as the date of their last expected visit.

The EXACT-PRO total score will be calculated by first summing the raw scores of all 14 items (score range: 0-51) and then looking up the corresponding EXACT-PRO total score in the table described in the Appendix 4 (converted score range: 0-100).

E-RS subdomain score is calculated as the sum from the relevant questions.

#### 16.2.1.2.2. **SGRQ**

St. George's Respiratory Questionnaire (SGRQ) is a questionnaire consisting of 17 questions, split into two parts. Part 1 consists of the first 8 questions and is related to the Symptoms subdomain. The remaining 9 questions are in Part 2, which are related to the Activity and Impacts subdomains. Each possible answer to each question has a weight assigned described in the Appendix 5.





Statistical Analysis Plan


Note that question 6 (How long did the worst respiratory attack last?) has an additional instruction, "Go to Question 7 if you did not have a severe attack". If question 6 has not been answered, it will be assigned a weight of zero.

#### Calculating the score

Subdomains:

- Symptoms items 1 to 8
- Activity items 11 and 15
- Impacts items 9, 10, 12, 13, 14, 16 and 17

The score for each component is calculated separately by dividing the summed weights by the maximum possible weight for that component and expressing the result as a percentage. It is not possible to have missing items in the questionnaire, as the data are collected in an electronic tablet which doesn't allow patients to skip between items.

 $Component\ score = 100* \frac{Sum\ of\ weights\ from\ all\ positive\ items\ in\ that\ component}{Sum\ of\ maximum\ weights\ for\ all\ items\ in\ that\ component}$ 

The total score is calculated similarly

 $Total\ score = 100* \frac{Sum\ of\ weights\ from\ all\ positive\ items\ in\ that\ questionnaire}{Sum\ of\ maximum\ weights\ for\ all\ items\ in\ that\ questionnaire}$ 

The higher the score the more severe impact of COPD on patient's life.

Sum of maximum possible weights for each component and Total:

Symptoms = 662.5

Activity = 1209.1

Impacts = 2117.8

Total = 3989.4

#### 16.2.1.2.3. **BDI/TDI**

Baseline Dyspnea Index (BDI) and Translational Dyspnea (TDI) are questionnaires that focus on three subdomains: Functional impairment, Magnitude of task and Magnitude of effort. BDI is collected at baseline (Day 1) and TDI is collected post-baseline (Weeks 6, 12 and 24).

Subdomain score is calculated as the sum from the related questions. Total score is calculated as the sum of the subdomain scores.





Statistical Analysis Plan


If at least one of the scores is missing, then total score is set to missing.

#### 16,2,1,3. Rescue Medications

Baseline use of rescue medication is the mean over the last 7 days of run-in phase, using only days where data was recorded:

# Sum of number of puffs taken days recorded

Use of medication per week is calculated as the mean use daily over 7 days, as described in the windowing conventions Section of the SAP, calculated only based on the days data was recorded/verified.

If less than 4 days of data are available for the week, the weekly mean is set to missing. If a patient discontinued then use study discontinuation end date, as the date of their last expected data input.

This will be documented as Albuterol/Salbutamol in the "Rescue Medication" page of the eCRF, as well as in the "Rescue Medication Use" diary entry.

The rescue medication use will be confirmed in the diary using the following rules:

- 1. If patient has put in rescue medication use then analyze as expected.
- If patient has not put in rescue medication use, then to confirm that there was no diary compliance issue, or IT issue, question "No Rescue Medication Confirmation" will be checked to make sure it is filled in correctly.
- 3. If patient has not put in rescue medication use and question "No Rescue Medication Confirmation" was not filled in correctly then this will be treated as diary compliance or IT issue and therefore this day will not be used as the day recorded for the weekly means calculation.

## 16.2.2. MISSING DATA METHODS FOR SECONDARY EFFICACY VARIABLES

## 16.2.2.1. MI method - continuous data

The analysis for key secondary endpoints (FEV $_1$  AUC $_{0-4h}$ , peak FEV $_1$ , morning trough FEV $_1$ , SGRQ total score and weekly mean E-RS total score) and for evening trough FEV1 and weekly rescue medication will be performed using MI based on the missing data assumption MAR. This process will follow four steps (below the example uses baseline FEV $_1$ , but it is repeated also for baseline of other key secondary endpoints mentioned above, excluding the ones evaluated weekly):





Statistical Analysis Plan


Partially impute the data for a monotone missing pattern with 100 as a number of imputations and "20905" as seed number. Employ the Markov Chain Monte Carlo (MCMC) method with treatment, region, background medication strata, smoking strata, baseline FEV<sub>1</sub> and <Visit data>. <Visit data> corresponds to all scheduled visits available for the parameter analyzed. Each visit will correspond to a covariate within the model.

#### The following SAS codes will be used:

```
proc mi data=<data1> out=<data2> nimpute=100 seed=20905;
   var <treatment> <region> <BackgroundMedStrata> <SmokingStrata>
   <baseline> <visits>;
   mcmc impute=monotone chain=multiple;
run:
```

2. Impute the monotone data using a regression imputation model. Apply by imputation using seed number "20905" with treatment, region, background medication strata, smoking strata, baseline FEV<sub>1</sub> and <Visit data>.

#### The following SAS codes will be used:

- 3. Each multiple imputed dataset in Step 2 will be analyzed separately, as described in Section 16.2.3 of the SAP.
- 4. The estimates (LS means, SE, CI and p-value) from the model analysis in Step 3 will be combined using Rubin's combination rules for statistical inference.

Note: For secondary endpoints that are evaluated weekly, the following updates will be implemented for the first 2 steps:

- 1. MI model will contain weekly means at all weeks available to impute the data to create a monotone missingness pattern, so will be imputed missing values at any week (i.e. Week 1, Week 2, ...).
- After this, the fully imputed dataset will include weekly means at weeks corresponding to scheduled visits in the MI model, and also only impute missing values at weeks corresponding to scheduled visits.





Statistical Analysis Plan


#### 16.2.2.2. MI method - binary data

For the analysis of proportion of SGRQ, weekly mean total E-RS and Morning trough  $FEV_1$  responders, an analysis will be performed using MI based on the missing data assumption MAR. This process will impute the continuous underlying data, as per 16.2.2.1 (morning trough  $FEV_1$ , SGRQ total score and weekly mean total E-RS), and then recalculate the binary outcome of responder or non-responder. The analysis will follow the steps below (Ratitch and O'Kelly, 2014, pp.124 - 127) (below the example uses morning trough  $FEV_1$ , but it is repeated also for other endpoints mentioned above):

- 1) Follow steps 1 and 2 from 16.2.2.1 for the continuous morning trough FEV<sub>1</sub> results.
- 2) For the imputed results re-calculate response, where a response is an improvement from baseline in morning trough  $FEV_1$  of 100 mL.
- 3) Analyse each multiply imputed dataset separately, as described in Section 16.2.3 of the SAP, producing LS Means, odd ratios and corresponding 95% confidence interval and p-value.
- 4) For the odds ratios:
  - a) Before applying Rubin's rule, apply a normalising transformation to the odds ratios as well as their standard errors. The distribution of the log of odds ratios approximates to a normal distribution. Therefore, calculate the transformed values, where OR is odds ratio, Lower/Upper CL are the confidence interval estimates of the ORs:

$$OR_{norm} = \log(OR)$$
 
$$SE_{norm} = \frac{(\log(Upper\ CL) - \log(Lower\ CL))}{(2 \times 1.96)}$$

- b) Appy Rubin's rule with PROC MIANALYZE to the transformed odds ratios with corresponding transformed standard errors.
- c) Back-transform the combined results as follows:

$$\begin{aligned} OR_{bt} &= exp^{OR_{norm}} \\ Lower\ CL_{bt} &= OR_{bt} \times e^{(-1.96 \times SE_{norm})} \\ Upper\ CL_{bt} &= OR_{bt} \times e^{(1.96 \times SE_{norm})} \end{aligned}$$

- 5) For the odds of response per treatment arm.
  - a) Take the LS means to be estimates of the log-odds of response per treatment arm and assume that they asymptotically tend to follow a normal distribution.
  - b) Appy Rubin's rule with PROC MIANALYZE to the LS means.
  - Transform the combined results by exponentiating to get the odds of response per treatment arm.



Statistical Analysis Plan


#### 16.2.2.3. MI method - range data

The sensitivity analysis for key secondary endpoints (SGRQ total score and weekly mean E-RS total score) and the main analysis of TDI will be performed using MI based on the missing data assumption MAR as described in the Section 16.2.2.1 of the SAP. Additionally, in the first 2 steps the MIN= and MAX= options will be used to restrict the possible values that can be drawn referred to each endpoint (Laura Rodwell, 2014).

#### 16.2.2.4. Other methods

As a sensitivity analysis, other missing data method for key secondary endpoints will follow the average imputation and tipping point approach taken for primary endpoint outlined in Section 16.1.2 of the SAP.

#### 16.2.3. ANALYSIS OF SECONDARY EFFICACY VARIABLES

#### 16.2.3.1. Change from baseline variables, incl. TDI

All variables used in change from baseline analysis (incl. average FEV<sub>1</sub> AUC<sub>0-4h</sub>, peak FEV<sub>1</sub>, morning trough FEV<sub>1</sub>, evening trough FEV<sub>1</sub>, mean weekly E-RS<sup>TM</sup>:COPD, SGRQ, mean weekly rescue medication and TDI) will be analyzed using ANCOVA approach, as described in Section 16.1.3 of the SAP. BDI will be used as a baseline for TDI. Missing data will be imputed using imputation described in Section 16.2.2 of the SAP. Continuous method will be used for lung function endpoints and the main analysis. Range method will be used for corresponding sensitivity analyses of SGRQ total score and weekly mean E-RS total score and the main analysis of TDI.

Model assumptions will be tested and solved, if failed, as per Section 16.1.3 of the SAP.

A plot of the mean change from baseline  $FEV_1$  to each post-dose  $FEV_1$  result over time will be created by subgroups of actual background medication strata and actual smoking strata, visit and treatment group.

A plot of the least squares means change from baseline to event over time will be presented (based on the ANCOVA analysis). Events will include weekly mean total E-RS score, SGRQ and weekly mean rescue medication use.

Only  $FEV_1$  measurements with BTR grades "Acceptable" and "Borderline Acceptable" are used in the analysis.



Copyright © 2009, 2010, 2012, 2016, 2018, 2019 IQVIA. All rights reserved. The contents of this document are confidential and proprietary to IQVIA Holdings Inc. and its subsidiaries. Unauthorized use, disclosure or reproduction is strictly prohibited.

Statistical Analysis Plan


#### 16.2.3.2. Proportion of SGRQ total responders

Proportion of responders, with an improvement from baseline in SGRQ total score of 4 or more will be analyzed using a logistic regression model with fixed effects for treatment, region, actual background medication strata and actual smoking strata at baseline and baseline SGRQ total score as covariate. Missing data will be imputed as described in Section 16.2.2.3 (range method).

## 16.2.4. SENSITIVITY ANALYSIS OF SECONDARY EFFICACY VARIABLES

For the key secondary endpoints the following sensitivity analysis will be performed at Week 12.

- Subgroup analysis as specified in Section 7.5 of the SAP.
- ANCOVA analysis with average imputation, as described in Section 16.1.2 of the SAP.
- ANCOVA analysis with MI, only considering baseline and Week 12 (for lung function parameters) in the imputation model, as described in Section 16.1.2 and 16.1.3 of the SAP.
- ANCOVA analysis with MI using the range data method as described in Section 16.2.2.3 for SGRQ total score and weekly mean total E-RS.
- Tipping point approach, as described in Section 16.1.2 of the SAP.
- Analysis with MI method, as described in Sections 16.2.2 and 16.2.3 of the SAP, based on PP population.
- For FEV<sub>1</sub> key secondary endpoints (FEV<sub>1</sub> AUC<sub>0-4h</sub>, peak FEV<sub>1</sub>, morning trough FEV<sub>1</sub>) additional sensitivity analysis will be performed:
  - MMRM model with treatment, visit and treatment by visit as fixed effect; baseline as
    covariate; patient as random factor; unstructured covariance by visit. If the model does
    not converge a compound symmetry covariance structure will be used. Kenward-Roger
    method will be used to estimate the model degrees of freedom.

- For weekly mean E-RS total score and SGRQ total score, additional analysis will be performed:
  - For weekly mean E-RS total score at 6, 12 and 24 weeks using ANCOVA approach, as described in Section  of the SAP, all patients with baseline mean = 0 will be excluded.
  - For SGRQ total score at 6, 12 and 24 weeks, using ANCOVA approach, as
    described in Section 16.2.3.1 of the SAP, all patients with baseline assessment done
    after dosing time and date will be excluded.

0



Statistical Analysis Plan


#### 16.3. OTHER EFFICACY

The other efficacy analyses will be performed for the mITT population.

- Moderate/severe COPD exacerbation frequency of patients using full study length, period truncated at week 24 visit and for patients in 48-week stratum (this individual study and pooled with data from study RPL554-CO-302).
- Time to first moderate/severe COPD exacerbation of patients using full study length, period truncated at week 24 visit and for patients in 48-week stratum (this individual study and pooled with data from study RPL554-CO-302).
- Study withdrawal before scheduled visit at 24 and 48 weeks.
- Change from baseline to post-baseline EQ-5D-5L using Health index and VAS score at Week 12
- HRU over 24 and 48 weeks
- Change from baseline FEV<sub>1</sub> to average FEV<sub>1</sub> AUC<sub>6-12h</sub> at Week 12
- E-RS responder analysis
- Morning trough FEV<sub>1</sub> responder analysis
- · Change from baseline SGRQ score by domain: symptoms, activity, impacts
- Change from baseline E-RS score by domain: breathlessness, cough and sputum, chest symptoms

#### 16.3.1. OTHER EFFICACY VARIABLES & DERIVATIONS

#### 16.3.1.1. COPD exacerbation

COPD exacerbations are collected on the "COPD Exacerbation" page of the eCRF and severity will be derived separately using data collected in the eCRF and as per the criteria specified in Section 11.6.1. of the study protocol.

Site must enter at least 2 major symptoms, or one major symptom and one minor symptom AND meet the severity criteria below, considered as a moderate/severe exacerbation of COPD.

The severity of the COPD exacerbation will be calculated as per the following:

**Moderate:** Worsening symptoms of COPD requiring a minimum of three days of treatment with oral/systemic corticosteroids and/ or antibiotics.

**Severe:** Worsening symptoms of COPD requiring in-patient hospitalization.



Statistical Analysis Plan


#### 16.3.1.2. Time to study withdrawal

Time to study withdrawal will be derived as follows:

- For patients who completed the study: Use the day of final week 24 or week 48 clinic visit, depending on which stratum the patient is randomized into
- For patients who did not complete the study but not lost to follow-up: If available, use the end of study date. If not available, use the last site contact out of any assessment (excluding eDiary).
- For patients who are lost to follow-up: the censoring date will be their last reported site contact.

#### 16.3.1.3. EQ-5D-5L

Quality of Life (QoL) was assessed using the EQ-5D-5L questionnaire. This questionnaire consits of 5 domains: mobility, self-care, usual activities, pain/discomfort and anxiety/depression with 5 possible responses from 1 (no problem) to 5 (unable). The sixth item, referred to as a visual analogue scale (VAS) score, is an index score to self-rate health from 0 (worst) to 100 (best). Each of the 5 domains will be summed through weighing system into a health index. The health index and VAS score will be analysed and listed and 5 domains will be only listed. It is not possible to have missing items in the questionnaire, as the data are collected in an electronic tablet which doesn't allow patients to skip between items. The weighting system is described in Appendix 6 of the SAP.

#### 16.3.1.4. HRU

HRU is measured by the following events: unscheduled visits to a physician office, visits to urgent care, visits to emergency department and hospitalizations for any cause and/or related to COPD and visits/contact due to COPD exacerbation. These will be recorded on the Log Form and "COPD Exacerbation" pages of the eCRF, respectively.

## 16.3.1.5. Patient Perception Survey

At the follow-up contact each patient will fill in a survey on their perception of what drug they were on. Data recorded on "Patient Perception Survey" page of the eCRF will be listed and summarized by treatment group for the following categories:

- Patients who correctly guessed their drug
- Patients who incorrectly guessed their drug
- · Patients who were unsure of their drug

#### 16.3.1.6. FEV1 AUC<sub>6-12h</sub>

Average FEV<sub>1</sub> AUC<sub>6-12h</sub> is calculated as described in Section 16.1.1.1 of the SAP.



Copyright © 2009, 2010, 2012, 2016, 2018, 2019 IQVIA. All rights reserved. The contents of this document are confidential and proprietary to IQVIA Holdings Inc. and its subsidiaries. Unauthorized use, disclosure or reproduction is strictly prohibited.

Statistical Analysis Plan


#### 16.3.1.7. E-RS total score responder

E-RS total score responder is defined as a decrease from baseline in the week mean total of E-RS score of greater than or equal to 2.

## 16.3.1.8. Morning trough FEV<sub>1</sub> responder

Morning trough  $FEV_1$  responder is defined as an increase from baseline in the Morning trough  $FEV_1$  greater than or equal to 100 mL.

#### 16.3.1.9. SGRQ domains

SGRQ questionnaire is composed of three domains: symptoms, activity, and impacts as described in Section 16.2.1.2.2 of the SAP. Subdomain scores are calculated as follows:

- Symptoms score = sum of items 1 to 8 of SGRQ questionnaire
- Activity score = sum of items 11 and 15 of SGRQ questionnaire
- Impacts score = sum of items 9, 10, 12, 13, 14, 16 and 17 of SGRQ questionnaire

#### 16,3,1,10, E-RS domains

E-RS EXACT-PRO questionnaire is composed of three domains: breathlessness, cough and sputum, and chest symptoms as described in Section 16.2.1.2.1 of the SAP. Scores are calculated as follows:

- Breathlessness score = sum of items 7 to 11 of E-RS questionnaire
- Cough and sputum score = sum of items 2 to 4 of E-RS questionnaire
- Chest symptoms score = sum of items 1, 5 and 6 of E-RS questionnaire

#### 16.3.2. MISSING DATA METHODS FOR OTHER EFFICACY VARIABLES

For EQ-5D-5L missing data will be imputed using imputation described in Section 16.2.2.13 of the SAP (MI range method) and FEV<sub>1</sub> AUC<sub>6-12h</sub> missing data, E-RS and SGRQ domain missing data will be imputed using imputation described in Section 16.2.2.1 of the SAP (MI continuous method). Morning trough FEV<sub>1</sub> responder missing data will be handled as described in Section **** of the SAP (MI range method). E-RS total score responder missing data will be imputed similar to the SGRQ total score responder analysis as described in Section 16.2.2.32 of the SAP (MI range method).

## 16.3.3. ANALYSIS OF OTHER EFFICACY VARIABLES

Change from baseline to average FEV<sub>1</sub> AUC<sub>6-12h</sub> will be analyzed using ANCOVA approach and missing data will be imputed using imputation, as described in Sections 16.1.3 and 16.2.2.1 of





Statistical Analysis Plan


the SAP, respectively.

Model assumptions will be tested and solved, if failed, as per Section 16.1.3 of the SAP.

The rate of and time to first moderate/severe COPD exacerbations will be analyzed in three cutoff rules:

- All patients (patients in 24-week and 48-week strata combined) using full study length
- Period truncated at Week 24 visit (patients in 24-week and 48-week strata combined)
- Patients in 48-week stratum using full study length

For each of the three rules above, the number of patients who experienced COPD exacerbation will be presented by week, follow-up and overall. Similarly, the duration of COPD exacerbation (in days) and the time in study will be calculated based on the cut-off rules.

Weekly percentage of patients who experienced COPD exacerbation will be based on the treatment population being analyzed. For All patients and Period truncated at Week 24 visit, the percentage will have denominator of mITT population. Analysis using 48-week stratum only will have mITT patients in this stratum as denominator.

For each cut-off rule, the number of moderate/severe COPD exacerbations will be analyzed using a negative binomial model adjusting for treatment, region, actual background medication strata and actual smoking strata, as well as using log study time (years) as an offset. If the model does not converge, the covariate that causes the issue will be removed from the model. The number of patients who experienced exacerbations and the number of exacerbations will also be presented using the data used to analyze negative binomial model.

The logic for time in study used as offset or for censoring purpose is as follows:

- For 24-week completers, use the day of final week 24 clinic visit. For 48-week completers, use the day of the final week 48 clinic visit.
- For non-completers who are not lost to follow-up, use the end of study date, which is assumed to be their end of study visit.
  - If no end of study date, use the last site contact out of any assessment (excluding eDiary)
- For subjects who are lost to follow-up, the censoring date will be at their last reported site contact.

Moderate/severe exacerbations occurring after the day used as offset will not be considered in the analysis. The treatment difference from the negative binomial model will be expressed as an





Statistical Analysis Plan


annualized risk ratio. The data will also be summarized by treatment group over duration of the study period. Only moderate/severe COPD exacerbations meeting the protocol-specified criteria will be presented in the listing.

Time to study medication withdrawal or study withdrawal will be presented per stratum and by the following subgroups: patients who withdrew from study medication/study before Week 24 visit and patients who withdrew from study medication/study before Week 48 visit for 48-week stratum.

Time to first moderate/severe COPD exacerbation during the study period will be presented for all patients using full study length, all patients using data truncated at week 24 visit, and patients in 48-week stratum. The primary analysis will include log-rank test stratified by region, actual background medication strata and actual smoking strata. Summary of number of patients with events and number of patients censored will be presented. Outcome will be visualized using a Kaplan-Meier plot.

The health index and VAS score for EQ-5D-5L questionnaire will be analyzed using ANCOVA approach, as described in Section 16.1.3 of the SAP, with data imputation described in Section 16.2.2.3 of the SAP.

HRU over a period truncated up to Week 24 visit for all patients (24-week and 48-week strata combined) and for 48-week stratum only will be summarized for each event and for overall count. HRU during follow-up period will not be presented.

- Sensitivity analysis or subgroup analysis may be considered following results of the
  patient perception survey. The survey will be summarized to investigate if there are any
  signs of breaching of the blind related to the appearance of study medication.
- Proportion of E-RS total score responders will be analyzed by means of a logistic regression model with fixed effects for treatment, region, actual background medication strata and actual smoking strata at baseline and baseline E-RS total score as covariate. Missing data will be imputed as described in Section 16.2.2.3 (range method).
- Proportion of responders, with an improvement from baseline in Morning trough FEV<sub>1</sub> of 100 mL or more will be analyzed using a logistic regression model with fixed effects for treatment, region, actual background medication strata and actual smoking strata at baseline and baseline Morning trough FEV<sub>1</sub> as covariate. Missing data will be imputed as described in Section 16.2.2.3 (range method).





Statistical Analysis Plan


 Change from baseline SGRQ scores and E-RS scores will be analyzed by domain using ANCOVA approach as described in Section 16.2.3.1 of the SAP.

#### 16.3.4. SENSITIVITY ANALYSIS OF OTHER EFFICACY VARIABLES

Sensitivity analysis with no data imputation, including only patients with data collected at the required visit while still on randomized treatment at scheduled visit, or at end of study visit within the visit window will be performed on the health index and VAS score for EQ-5D-5L questionnaire and analyzed using ANCOVA approach, as described in Section 16.1.3 of the SAP.

For E-RS total score responder analysis a sensitivity analysis using other approaches MI imputation using the continuous data method described in Section 16.2.2.1.

Sensitivity analysis for time to first moderate/severe COPD exacerbation will be done for the three data groups used in the main analysis: all patients, period truncated at week 24 visit, and patients in 48-week stratum, as described in Section 16.3.3 of the SAP. The analysis will be done using Cox proportional hazards regression model stratified by region, background medication strata and smoking strata. Patients without exacerbations will be censored (as described in the logic for time in study above) at last day in the treatment period, including period of recording after possible treatment withdrawal. Moderate/severe COPD exacerbations that happened in the follow-up period will be excluded from the analysis since these occur after censoring. The treatment difference in the Cox model will be expressed as a hazard ratio.

Testing proportional hazard assumptions:

- Check that the covariates are independent of each other through proc phreg in SAS software.
- 2. Check that the hazard (hazard ratio) is independent of time through log(-log(survival)) vs log(time) plot and an interaction test for treatment times log(time).

#### 16.4. EVALUATION INCLUDING EXCLUDED SITES

Sites were removed from the mITT. As a check of the impact of this exclusion the following analyses will be performed in the Extended mITT population.



Copyright © 2009, 2010, 2012, 2016, 2018, 2019 IQVIA. All rights reserved. The contents of this document are confidential and proprietary to IQVIA Holdings Inc. and its subsidiaries. Unauthorized use, disclosure or reproduction is strictly prohibited.

Statistical Analysis Plan


- Analysis of FEV<sub>1</sub> AUC<sub>0-12</sub>
- Analysis of peak FEV<sub>1</sub>
- Analysis of E-RS total score
- · Analysis of SGRQ total score
- Analysis of morning trough FEV<sub>1</sub>
- Responder analysis of SGRQ total score

## 17. SAFETY OUTCOMES

All outputs for safety outcomes will be based on the SAF set.

There will be no statistical comparisons between the treatment groups for safety data, unless otherwise specified with the relevant section.

## 17.1. ADVERSE EVENTS

Adverse Events (AEs) will be coded using MedDRA central coding dictionary. The version of MedDRA to be used will be specified prior to database lock.

Treatment-emergent adverse events (TEAEs) are defined as AEs that started or worsened in severity on or after the first dose of study medication. Laboratory or ECG findings from procedures or samples drawn prior to the first does of study medication that are assessed/overread after randomization will be considered pre-treatment.

In the case where it is not possible to define an AE as treatment-emergent or not, the AE will be classified by the worst case; i.e. treatment-emergent.

See Appendix 2 for handling of partial dates for AEs.

An overall summary of number of patients within each of the categories described in the subsection below, will be provided as specified in the shells. The summary AE tables will be presented for overall (up to the end of study for all patients) and separately for data up to week 24 visit (regardless of which treatment duration stratum a patient is randomized into) and data from week 24 up to week 48 visit.

In addition, the number of patients with each of the following AE events will be presented by SOC and PT and summarized by treatment group and different period (i.e. Treatment period (+3





Statistical Analysis Plan


days), Follow-up (last dose + 4 days) and Overall). These will also be presented for overall, up to week 24 visit, and from week 24 up to week 48 visit:

- TEAE
- · TEAEs causally related to study medication
- Serious TEAEs
- · TEAEs with an outcome of death
- · TEAEs leading to discontinuation of blinded study medication
- TEAEs leading to withdrawal from study (TEAEs with a diagnosis of COVID-19, TEAEs with no diagnosis of COVID-19)
- TEAEs by maximum severity (Mild, Moderate, Severe)

AEs will be identified by using the "Adverse Events" page of the eCRF. Listings will include TEAEs and Non-TEAEs.

Treatment period is defined as the period from the date and time of first dose up to the last date and time of last dose.

Follow-up is defined as the period from after the date and time of last dose up to the last date recorded on the study.

#### 17.1.1. ALL TEAES

Incidence of TEAEs will be presented by SOC and PT and broken down further by maximum severity and relationship to study medication.

#### 17.1.1.1. Severity

Severity is classed as mild/ moderate/ severe (increasing severity). TEAEs starting after the first dose of study medication with a missing severity will be classified as severe. If patient reports a TEAE more than once within that SOC/ PT, the AE with the worst-case severity will be used in the corresponding severity summaries.

## 17.1.1.2. Relationship to Study Medication

Relationship, as indicated by the Investigator, is classed as "unknown", "unrelated", "unlikely to be related", "possibly related" and "probably related" (increasing probability of relationship). A "related" TEAE is defined as a TEAE with a relationship to study medication as "possibly related" or "probably related" to study medication. TEAEs with a missing relationship to study medication will be regarded as "probably related" to study medication. If a patient reports the same AE more than once within that SOC/PT, the AE with the worst case relationship to study medication will be used in the corresponding relationship summaries.





Statistical Analysis Plan


#### 17.1.2. TEAES LEADING TO DISCONTINUATION OF STUDY MEDICATION

TEAEs leading to discontinuation of study medication are AEs recorded as "Study Treatment Permanently Discontinued" on the "Adverse Events" page of the eCRF.

For TEAEs leading to discontinuation of study medication, summaries of incidence rates (frequencies and percentages) by SOC and PT will be prepared.

#### 17.1.3. SERIOUS ADVERSE EVENTS

Serious adverse events (SAEs) are those events recorded as "Serious" on the "Adverse Events" page of the eCRF. A summary of serious TEAEs by SOC and PT and by treatment group and different period (i.e. Treatment period, Follow-up and Overall) will be prepared.

#### 17.1.4. ADVERSE EVENTS LEADING TO DEATH

TEAEs leading to Death are those events which are recorded as "Fatal" on the "Adverse Events" page of the eCRF. A summary of TEAEs leading to death by SOC and PT will be prepared.

#### 17.2. LABORATORY EVALUATIONS

Results from the central laboratory (or local laboratory where this is required) will be included in the reporting of this study for chemistry, hematology and viral serology. A list of laboratory assessments to be included in the outputs is included in the Appendix 3 of the study protocol. The handling of Russian laboratories is detained in Section 6.10 of the SAP.

Presentations of all laboratory tests will use either conventional or standard international (SI) units. However, certain laboratory tests will also be presenting using US units, including liver tests. Laboratory evaluations will be presented separately for 24-week and 48-week strata.

The handling of re-test and unscheduled measurements is detailed in Section 6.4 of the SAP.

The following summaries will be provided for chemistry and hematology data:

- Actual and change from baseline by visit (for quantitative measurements)
- · Incidence of abnormal values according to normal range criteria
- Shift from baseline according to normal range criteria (for quantitative measurements and categorical measurements)
- Shift from baseline according to markedly abnormal criteria (for quantitative measurements and categorical measurements)
- · Listing of patients meeting markedly abnormal criteria



Statistical Analysis Plan


Viral serology, COVID-19 sample, chemistry and hematology will be listed. The original reference ranges recorded by the local sites or provided by InVitro used for chemistry and hematology parameters will be included in the listing.

## 17.2.1. LABORATORY REFERENCE RANGES AND CLINICALLY SIGNIFICANT ABNORMAL CRITERIA

Quantitative laboratory measurements will be compared with the relevant laboratory reference ranges in SI units and categorized as:

- Low: Below the lower limit of the laboratory reference range.
- Normal: Within the laboratory reference range (upper and lower limit included).
- High: Above the upper limit of the laboratory reference range.

In addition to the high and low quantitative laboratory assignments (as identified by means of the laboratory reference ranges), clinically significant abnormal quantitative chemistry laboratory assessments will also be identified in accordance with the predefined markedly abnormal criteria as presented in Table 4.

If ULN or LLN have " $\leq$ X" or " $\geq$ X" then "X" will be used for analysis and " $\leq$ X" or " $\geq$ X" will only be used in listings.

Table 4: Clinically Significant abnormal criteria for laboratory parameters

| Parameter | Clinically Significant Abnormally High Criteria |
|---|---|
| Alanine Aminotransferase (ALT) | > 3 times Upper Limit of Normal Range |
| Alkaline Phosphatase | > 3 times Upper Limit of Normal Range |
| Aspartate Aminotransferase (AST) | > 3 times Upper Limit of Normal Range |
| Creatinine | >221 μmol/L |
| Gamma Glutamyltransferase (GGT) | > 3 times Upper Limit of Normal Range |
| Total Bilirubin | > 3 times Upper Limit of Normal Range |

#### 17.3. ECG EVALUATIONS

Results from the central Electrocardiogram (ECG) Reading Centre will be included in the





Statistical Analysis Plan


reporting of this study. ECG evaluations will be presented separately for 24-week and 48-week strata.

The following ECG parameters will be reported for this study:

- PR Interval (msec)
- QRS Interval (msec)
- QT Interval (msec)
- QTcF Interval (msec)
- QTcB Interval (msec)
- Heart Rate (beats per minute [bpm])
- Overall assessment of ECG (Investigator's judgment):
  - Normal
  - o Abnormal, Not Clinically Significant (ANCS)
  - o Abnormal, Clinically Significant (ACS)

On Day 1, prior to dosing, triplicate ECGs must be performed. Triplicate results will be used in the summaries by taking an average of the 3 results. The average of the 3 results will be the baseline. Baseline for the investigator's judgement will be the mode judgment of the 3 results. In the case of multiple modes, the mode with the worst-case judgment (Normal<ANCS<ACS) will be used as baseline.

If only 2 ECG measurements instead of triplicate on Day 1 pre-dose, take average of the two; if only 1 measurement then this will be the baseline.

The handling of re-test and unscheduled measurements is detailed in Section 6.3 of the SAP.

If there were more measurements on a scheduled visit, choose measurement as follows:

- 1. Choose first triplicate, if more than one done.
- 2. If done on Day 1, ensure you choose measurement that it is prior to dosing.
- If there are more than 1 ECG measurements, choose the scheduled one where interpretation of the measurement from the vendor data is not "UNABLE TO EVALUATE".
  - a. If pre-dose/post-dose and interpretation of the measurement from the vendor data is "UNABLE TO EVALUATE" and no further pre-dose/post-dose unscheduled visits on the same day, respectively set to missing
  - b. If pre-dose/post-dose and interpretation of the measurement from the vendor data is "UNABLE TO EVALUATE" and there is another unscheduled pre-dose/post-dose choose next unscheduled visit on the same day



Statistical Analysis Plan


The following summaries will be provided for ECG data:

- Actual and change from baseline by visit (for quantitative measurements)
- Shift table representing changes from Normal, ANCS and ACS, using Investigator's judgement
- Incidence of markedly abnormal criteria
- · Listing of patients meeting markedly abnormal criteria

#### 17.3.1. ECG MARKEDLY ABNORMAL CRITERIA

Markedly abnormal quantitative ECG measurements will be identified in accordance with the following predefined markedly abnormal criteria:

- Absolute values for QT interval, QTcB interval and QTcF interval will be classified as:
  - o > 450 msec
  - o > 480 msec
  - o > 500 msec
- Change from Baseline for QT interval, QTcB interval and QTcF will be classified as:
  - >30 msec increase from baseline
  - o >60 msec increase from baseline

#### 17.4. VITAL SIGNS

The following Vital Signs measurements will be reported for this study:

- Supine Systolic Blood Pressure (mmHg)
- Supine Diastolic Blood Pressure (mmHg)
- Supine Pulse Rate (bpm)
- Respiratory Rate (breaths/min)
- Temperature (° C)
- Body weight (kg)
- Height (cm)
- BMI (kg/m<sup>2</sup>)

Vital signs will be presented separately for 24-week and 48-week strata. The following summaries will be provided for vital signs data (excluding respiratory rate, temperature, body weight, height and BMI):

- · Actual and change from baseline by visit
- Incidence of markedly abnormal values



Statistical Analysis Plan


- · Shift from baseline according to markedly abnormal criteria
- · Listing of patients meeting markedly abnormal criteria

Respiratory rate, temperature, body weight, height and BMI will be listed.

#### 17.4.1. VITAL SIGNS MARKEDLY ABNORMAL CRITERIA

Markedly abnormal quantitative Vital Signs measurements will be identified in accordance with the predefined markedly abnormal criteria found in Table 5.

Markedly Abnormal Post-Baseline Vital Signs

| Variable | Unit | Abnormally Low | Abnormally High |
|---|---|---|---|
| SBP | mmHg | <ul> <li>A decrease from<br/>Baseline of ≥40</li> <li>Value ≤90</li> </ul> | - An increase from Baseline of<br>≥40<br>- Value ≥180 |
| DBP | mmHg | <ul> <li>A decrease from<br/>Baseline of ≥20</li> <li>Value ≤50</li> </ul> | <ul> <li>An increase from<br/>Baseline of ≥20</li> <li>Value ≥105</li> </ul> |
| Pulse rate | Bpm | <ul> <li>A decrease from<br/>Baseline of ≥30</li> <li>Value ≤50</li> </ul> | <ul> <li>An increase from<br/>Baseline of ≥30</li> <li>Value ≥110</li> </ul> |

## 17.5. COVID-19

From study initiation until 5Nov2021, patients with positive COVID-19 test indicating an active COVID-19 infection were withdrawn from the study.

A protocol clarification letter dated 5Nov2021 clarified that active infection includes known symptoms of COVID-19.

A protocol clarification letter dated 21Apr2022 clarified that active infection includes known lower respiratory symptoms of COVID-19.

Patients who discontinued due to COVID-19 will be summarized in the disposition table. Data collected on the "COVID-19 Visit Impact" eCRF page will be summarized by visit. Data on the optional COVID-19 testing will be listed.





Statistical Analysis Plan


## 17.6. PNEUMONIA

Pneumonia details recorded in the "Pneumonia" page of the eCRF will be listed.

## 17.7. EVALUATION INCLUDING EXCLUDED SITES

The following analyses will be performed on the Extended Safety Set:

- · Summary of TEAEs
- TEAEs by SOC and PT
- Related TEAEs by SOC and PT
- · Serious TEAEs by SOC and PT
- · Markedly abnormal values for selected chemistry parameters
- · Markedly abnormal values for vital signs
- Markedly abnormal values for ECG parameters

## 18. DATA NOT SUMMARIZED OR PRESENTED

The other variables and/or domains not summarized or presented are:

- Comments
- · Physical Examinations, as it is not collected within eCRF

These domains and/or variables will not be summarized or presented, but if collected will be available in the clinical study database, SDTM and/or ADaM datasets.





Statistical Analysis Plan


## 19. REFERENCES

Devlin N, S. K. (2017, June). Valuing health-related quality of life: An EQ-5D-5L value set.

EMA. (2014, October). *EXACT-PRO Initiative*. Retrieved from http://www.ema.europa.eu/docs/en\_GB/document\_library/Other/2015/04/WC500185444.pdf

EQ-5D. (2019, September). EQ-5D-5L User Guide v3.0. Retrieved from EQ-5D.

Golicki D, J. M. (2019, June). Valuation of EQ-5D-5L Health States in Poland: the First EQ-VT-Based.

ICH. (2019). ADDENDUM ON ESTIMANDS AND SENSITIVITY ANALYSIS IN CLINICAL TRIALS.

Jones, P. P. (2009, June). ST GEORGE'S RESPIRATORY QUESTIONNAIRE MANUAL.

Laura Rodwell, K. J. (2014). Comparison of methods for imputing limited-range variables: a simulation study. *BMC Medical Research Methodology*.

Merinopoulou E, R.-C. M. (2016). COPD exacerbations by disease severity in England. *Int J Chron Obstruct Pulmon Dis.* 

Pickard S, L. E. (2019, August). United States Valuation of EQ-5D-5L Health States Using an International.

Ratitch B., O. M. (2014). Clinical Trials with Missing Data: A Guide for Practitioners. John Wiley & Sons, Ltd.

SAS Institute, Inc. (1999). SAS Procedures Guide, version 8. Cary, NC: SAS Institute.



Statistical Analysis Plan


## APPENDIX 1. Programming Conventions for Outputs

## **DATES & TIMES**

Depending on data available, dates and times will take the form yyyy-mm-ddThh:mm:ss.

## SPELLING FORMAT

English US.

## PRESENTATION OF TREATMENT GROUPS

For outputs, treatment groups will be represented as follows and in the given order:

| Treatment Group | For Tables, Listings and Graphs |
|-----------------|---------------------------------|
| Ensifentrine | Ensifentrine |
| Placebo | Placebo |
| Not Randomized | Not Randomized |

## DECIMAL PLACES

The decimal places for this study will use the following rules, unless otherwise stated.

Value = x dp

Mean = x+1 dp

Standard Deviation = x+2 dp

Median = x+1 dp

Q1/Q3 = x+1 dp

Minimum/Maximum = x dp

CI = x+1 dp

In case a variable has values with infinite decimal places, the following rules will be used:

Value = 1 dp

Mean = 2 dp

Standard Deviation = 3 dp

Median = 2 dp

Q1/Q3 = 2 dp

Minimum/Maximum = 1 dp




Statistical Analysis Plan


CI = 2 dp

For spirometry data we will present outputs with decimal places for value as follows:

- Values in liters = 3 dp, i.e. mean/median/Q1/Q3/CI in liters = 4 dp, standard deviation = 5 dp and minimum/maximum = 3 dp.
- Values in milliliters = 0 dp, i.e. mean/median/Q1/Q3/CI in liters = 1 dp, standard deviation = 2 dp and minimum/maximum = 0 dp.
- Percentage values = 1 dp, i.e. mean/median/Q1/Q3/CI in liters = 2 dp, standard deviation = 3 dp and minimum/maximum = 1 dp.

P-values will be presented to 4dp.

#### PRESENTATION OF VISITS

For outputs, visits will be represented as follows and in that order:

| Long Name (default) | Short Name |
|---------------------|------------|
| Screening | Screening |
| day 1 | day 1 |
| week 6 | week 6 |
| week 12 | week 12 |
| week 18 | week 18 |
| week 24 | week 24 |
| week 30 | week 30 |
| week 36 | week 36 |
| week 42 | week 42 |
| week 48 | week 48 |
| Follow-up | Follow-up |

#### LISTINGS

All listings will be ordered by the following (unless otherwise indicated in the template):





Statistical Analysis Plan


- Randomized treatment group (or treatment received if it's a safety output), first by active
  dose and then placebo,
- · Center-patient ID,
- · Date and time (where applicable),
- For listings where non-randomized patients are included, these will appear in a category after the randomized treatment groups labeled 'Not Randomized'.

#### **TABLES**

All tables presenting multiple events that map to a SOC and PT will be counted only once, per unique patient, for incidence counts. Events will be presented in descending frequency of SOC and PT (unless otherwise indicated in the shells).



Statistical Analysis Plan


#### APPENDIX 2. PARTIAL DATE CONVENTIONS

Imputed dates will NOT be presented in the listings.

#### ALGORITHM FOR TREATMENT EMERGENCE OF ADVERSE EVENTS:

| START DATE | STOP DATE | ACTION |
|---|---|---|
| Known | Known/Partial/<br>Missing | If start date < study med start date, then not TEAE If start date >= study med start date, then TEAE |
| Partial, but known components show that it cannot be on or after study med start date | Known/Partial/<br>Missing | Not TEAE |
| Partial, could be on or<br>after study med start<br>date<br>OR Missing | Known | If stop date < study med start date, then not TEAE If stop date >= study med start date, then TEAE |
| | Partial | Impute stop date as latest possible date (i.e. last day of month if day unknown or 31st December if day and month are unknown), then: If stop date < study med start date, then not TEAE If stop date >= study med start date, then TEAE |
| | Missing | Assumed TEAE |





Statistical Analysis Plan


#### ALGORITHM FOR PRIOR/PRIOR CONCOMITANT / CONCOMITANT MEDICATIONS:

| START | STOP | ACTION |
|---|---|---|
| DATE | DATE | |
| Known | Known | If stop date < study med start date, assign as prior If stop date >= study med start date and start date < study med start, assign as prior concomitant If stop date >= study med start date and (start date > study med start or start date <= end of treatment), assign as concomitant If start date > end of treatment, assign as post study |
| | Partial | Impute stop date as latest possible date (i.e. last day of month if day unknown or 31st December if day and month are unknown), then: If stop date < study med start date, assign as prior If stop date >= study med start date and start date < study med start, assign as prior concomitant If stop date >= study med start date and (start date > study med start or start date <= end of treatment), assign as concomitant If start date > end of treatment, assign as post study |
| | Missing | If stop date is missing could never be assumed a prior medication If stop date >= study med start date and start date < study med start, assign as prior concomitant If stop date >= study med start date and (start date > study med start or start date <= end of treatment), assign as concomitant If start date > end of treatment, assign as post study |







Statistical Analysis Plan 

| STOP | ACTION |
|---|---|
| DATE | |
| Known | Impute start date as earliest possible date (i.e. first day of month if day unknown or 1st January if day and month are unknown), then: If stop date < study med start date, assign as prior If stop date >= study med start date and start date < study med start, assign as prior concomitant If stop date >= study med start date and (start date > study med start or start date <= end of treatment), assign as concomitant If start date > end of treatment, assign as post study |
| Partial | Impute start date as earliest possible date (i.e. first day of month if day unknown or 1st January if day and month are unknown) and impute stop date as latest possible date (i.e. last day of month if day unknown or 31st December if day and month are unknown), then: If stop date < study med start date, assign as prior If stop date >= study med start date and start date < study med start, assign as prior concomitant If stop date >= study med start date and (start date > study med start or start date <= end of treatment), assign as concomitant If start date > end of treatment, assign as post study |
| Missing | Impute start date as earliest possible date (i.e. first day of month if day unknown or 1st January if day and month are unknown), then: If stop date is missing could never be assumed a prior medication If stop date >= study med start date and start date < study med start, assign as prior concomitant If stop date >= study med start date and (start date > study med start or start date <= end of treatment), assign as concomitant If start date > end of treatment, assign as post study |
| | Partial |





Statistical Analysis Plan


| START<br>DATE | STOP<br>DATE | ACTION |
|---|---|---|
| Missing | Known | If stop date < study med start date, assign as prior If stop date >= study med start date, assign as concomitant Cannot be assigned as 'prior concomitant' and 'post treatment' |
| | Partial | Impute stop date as latest possible date (i.e. last day of month if day unknown or 31st December if day and month are unknown), then: If stop date < study med start date, assign as prior If stop date >= study med start date, assign as concomitant Cannot be assigned as 'prior concomitant' and 'post treatment' |
| | Missing | Assign as concomitant |

Statistical Analysis Plan 

#### **ALGORITHM FOR CONCOMITANT ILLNESSES:**

| START | STOP | ACTION |
|---|---|---|
| DATE | DATE | |
| Known | Known | If stop date > date of first treatment dose and start date <= date |
| | | of first treatment dose, assign as concomitant illness |
| | Partial | Impute stop date as latest possible date (i.e. last day of month if |
| | | day unknown or 31st December if day and month are |
| | | unknown), then: |
| | | If stop date > date of first treatment dose and start date <= date |
| | 2.61 | of first treatment dose, assign as concomitant illness |
| | Missing | If stop date is missing then assume concomitant illness |
| Partial | Known | Impute start date as earliest possible date (i.e. first day of month |
| | | if day unknown or 1st January if day and month are unknown), |
| | | then: |
| | | If stop date > date of first treatment dose and start date <= date of first treatment dose, assign as concomitant illness |
| | Partial | Impute start date as earliest possible date (i.e. first day of month |
| | | if day unknown or 1st January if day and month are unknown) |
| | | and impute stop date as latest possible date (i.e. last day of |
| | | month if day unknown or 31st December if day and month are |
| | | unknown), then: |
| | | If stop date > date of first treatment dose and start date <= date |
| | 3.00 | of first treatment dose, assign as concomitant illness |
| | Missing | Impute start date as earliest possible date (i.e. first day of month |
| | | if day unknown or 1st January if day and month are unknown), then: |
| | | If stop date is missing then assume concomitant illness |
| | | if stop date is missing their assume concomitant finiess |
| Missing | Known | If stop data > data of first treatment dose assign as concemitant |
| Missing | Kilowii | If stop date > date of first treatment dose, assign as concomitant illness |





Statistical Analysis Plan


| START<br>DATE | STOP<br>DATE | ACTION |
|---|---|---|
| | Partial | Impute stop date as latest possible date (i.e. last day of month if day unknown or 31st December if day and month are unknown), then: If stop date > date of first treatment dose, assign as concomitant illness |
| | Missing | If stop date is missing then assume concomitant illness |



Statistical Analysis Plan 

#### APPENDIX 3. ANNOTATED EXACT FOR RAW SCORE ASSIGNMENT

| 1. Did your chest feel congested today? | 0.Not at all |
|---|---|
| | 1.Slightly |
| | 2.Moderately |
| | 3.Severely |
| | 4.Extremely |
| 2. How often did you cough today? | 0.Not at all |
| | 1.Rarely |
| | 2.Occasionally |
| | 3.Frequently |
| | 4.Almost constantly |
| 3. How much mucus (phlegm) did you bring up when | 0.None at all |
| coughing today? | 1.A little |
| | 1.Some |
| | 2.A great deal |
| | 3.A very great deal |
| 4. How difficult was it to bring up mucus (phlegm) | 0.Not at all |
| today? | 1.Slightly |
| | 2.Moderately |
| | 3.Quite a bit |
| | 4.Extremely |
| 5. Did you have chest discomfort today? | 0.Not at all |
| | 1.Slight |
| | 2.Moderate |
| | 3.Severe |
| | 4.Extreme |
| 6. Did your chest feel tight today? | 0.Not at all |
| | 1.Slightly |
| | 2.Moderately |
| | 3.Severely |
| | 4.Extremely |
| 7. Were you breathless today? | 0.Not at all |
| | 1.Slightly |
| | 2.Moderately |
| | 3.Severely |
| | 4.Extremely |
| 8.Describe how breathless you were today | 0.Unaware of breathlessness |





Statistical Analysis Plan 

| | 1.Breathless during strenuous activity |
|---|---|
| | 2.Breathless during light activity |
| | 3.Breathless when washing or dressing |
| | 3.Present when resting |
| 9. Were you short of breath today when performing | 0.Not at all |
| your usual personal care activities like washing or | 1.Slightly |
| dressing? | 2.Moderately |
| | 3.Severely |
| | 3.Extremely |
| | 4.Too breathless to do these |
| 10. Were you short of breath today when performing | 0.Not at all |
| your usual indoor activities like cleaning or household | 1.Slightly |
| work? | 2.Moderately |
| | 3.Severely |
| | 3.Extremely |
| | 3.Too breathless to do these |
| 11. Were you short of breath today when performing | 0.Not at all |
| your usual activities outside the home such as yard | 1.Slightly |
| work or errands? | 2.Moderately |
| | 3.Severely |
| | 3.Extremely |
| | 3.Too breathless to do these |
| 12. Were you tired or weak today? | 0.Not at all |
| | 1.Slightly |
| | 2.Moderately |
| | 3.Severely |
| | 4.Extremely |
| 13. Last night, was your sleep disturbed? | 0.Not at all |
| | 1.Slightly |
| | 2.Moderately |
| | 3.Severely |
| | 4.Extremely |
| 14. How scared or worried were you about your lung | 0.Not at all |
| problems today? | 1.Slightly |
| • | 2.Moderately |
| | 3.Severely |
| | 3.Extremely |
| | J.EAUCHICIY |

Statistical Analysis Plan


# APPENDIX 4. RAW SUMMED SCORE TO SCALE CONVERSION TABLE FOR EXACT TOTAL SCORE

| Raw Summed | EXACT Total | Raw Summed | EXACT Total |
|------------|-------------|------------|-------------|
| Score | Score | Score | Score |
| 0 | 0 | 26 | 50 |
| 1 | 8 | 27 | 51 |
| 2 | 13 | 28 | 52 |
| 3 | 17 | 29 | 53 |
| 4 | 20 | 30 | 54 |
| 5 | 23 | 31 | 55 |
| 6 | 25 | 32 | 57 |
| 7 | 27 | 33 | 58 |
| 8 | 28 | 34 | 59 |
| 9 | 30 | 35 | 60 |
| 10 | 31 | 36 | 61 |
| 11 | 33 | 37 | 63 |
| 12 | 34 | 38 | 64 |
| 13 | 36 | 39 | 65 |
| 14 | 37 | 40 | 67 |
| 15 | 38 | 41 | 68 |
| 16 | 39 | 42 | 70 |
| 17 | 40 | 43 | 72 |
| 18 | 41 | 44 | 73 |
| 19 | 42 | 45 | 75 |
| 20 | 43 | 46 | 77 |
| 21 | 44 | 47 | 80 |
| 22 | 46 | 48 | 83 |
| 23 | 47 | 49 | 87 |
| 24 | 48 | 50 | 92 |
| 25 | 49 | 51 | 100 |





Statistical Analysis Plan 

### APPENDIX 5. SGRQ ITEM WEIGHTS

| Question | Answers | Weight |
|---|---|---|
| Part 1 | | |
| Question 1: Over the past 4 weeks, I have | | |
| coughed | Almost every day | 80.6 |
| | Several days a week | 63.2 |
| | A few days a month | 29.3 |
| | Only with respiratory infections | 28.1 |
| | Not at all | 0.0 |
| Question 2: Over the past 4 weeks, I have | | |
| brought up phlegm (sputum) | Almost every day | 76.8 |
| | Several days a week | 60.0 |
| | A few days a month | 34.0 |
| | Only with respiratory infections | 30.2 |
| | Not at all | 0.0 |
| Question 3: Over the past 4 weeks, I have | | |
| shortness of breath | Almost every day | 87.2 |
| | Several days a week | 71.4 |
| | A few days a month | 43.7 |
| | Only with respiratory infections | 35.7 |
| | Not at all | 0.0 |
| Question 4: Over the past 4 weeks, I have | | |
| wheezing attacks | Almost every day | 86.2 |
| | Several days a week | 71.0 |
| | A few days a month | 45.6 |
| | Only with respiratory infections | 36.4 |
| | Not at all | 0.0 |
| Question 5: How many times during the | | |
| past 4 weeks have you suffered from | More than 3 times | 86.7 |
| severe or very unpleasant respiratory | 3 times | 73.5 |
| attacks? | 2 times | 60.3 |
| | 1 time | 44.2 |
| | None of the time | 0.0 |
| Question 6: How long did the worst | | 10 mm m m m m m m m m m m m m m m m m m |
| respiratory attack last? | A week or more | 89.7 |
| (Go to Question 7 if you did not have a | 3 or more days | 73.5 |
| severe attack) | 1 or 2 days | 58.8 |

Statistical Analysis Plan


| | Less than a day | 41.9 |
|---|---|---|
| Question 7: Over the past 4 weeks, in a | | |
| typical week, how many good days (with | No good days | 93.3 |
| few respiratory problems) have you had? | 1 or 2 good days | 76.6 |
| | 3 or 4 good days | 61.5 |
| | Nearly every day was good | 15.4 |
| | Every day was good | 0.0 |
| Question 8: If you wheeze, is it worse | | |
| when you get up in the morning? | No | 0.0 |
| | Yes | 62.0 |
| Part 2 | | |
| Question 9: How would you describe your | | |
| respiratory condition? | The most important problem I have | 83.2 |
| <del>-</del> | Causes me quite a lot of problems | 82.5 |
| | Causes me a few problems | 34.6 |
| | Causes no problem | 0.0 |
| Question 10: If you ever held a job | • | |
| , | My respiratory problems made me | 88.9 |
| | stop working altogether | 3846.3380.794 |
| | My respiratory problems interfere | 77.6 |
| | with my job or made me change my | AN RESTOCUES AND |
| | job | |
| | My respiratory problems do not affect | 0.0 |
| | my job | |
| Question 11: Questions about what | | |
| activities usually make you short of breath | Sitting or lying still | 90.6 |
| these days | Washing or dressing yourself | 82.8 |
| | Walking around the house | 80.2 |
| | Walking outside on level ground | 81.4 |
| | Walking up a flight of stairs | 76.1 |
| | Walking up hills | 75.1 |
| | Playing sports or other physical | 72.1 |
| | activities | |
| Question 12: More questions about your | | 6 |
| cough and shortness of breath these days | Coughing hurts | 81.1 |
| | Coughing makes me tired | 79.1 |
| | I am short of breath when I talk | 84.5 |
| | I am short of breath when I bend over | 76.8 |



Statistical Analysis Plan 

| | My coughing or breathing disturbs my sleep | 87.9 |
|---|---|---|
| | I get exhausted easily | 84.0 |
| Question 13: Questions about other effects your respiratory problems may | | |
| have on you these days | My cough or breathing is embarrassing in public | 74.1 |
| | My respiratory problems are a<br>nuisance to my family, friends or<br>neighbors | 79.1 |
| | I get afraid or panic when I cannot catch my breath | 87.7 |
| | I feel that I am not in control of my respiratory problems | 90.1 |
| | I do not expect my respiratory<br>problems to get any better | 82.3 |
| | I have become frail or an invalid<br>because of my respiratory problems | 89.9 |
| | Exercise is not safe for me | 75.7 |
| | Everything seems too much of an effort | 84.5 |
| Question 14: Questions about your | | |
| respiratory treatment | My treatment does not help me very much | 88.2 |
| | I get embarrassed using my<br>medication in public | 53.9 |
| | I have unpleasant side effects from my medication | 81.1 |
| | My treatment interferes with my life a lot | 70.3 |
| Question 15: Questions about how | | |
| activities may be affected by your respiratory problems | I take a long time to get washed or dressed | 74.2 |
| | I cannot take a bath or shower, or I take a long time | 81.0 |
| | I walk more slowly than other people, or I stop to rest | 71.7 |





Statistical Analysis Plan 

| | Jobs such as housework take a long | 70.6 |
|---|---|---|
| | time, or I have to stop to rest | |
| | If I walk up one flight of stairs, I have | 71.6 |
| | to go slowly or stop | |
| | If I hurry or walk fast, I have to stop | 72.3 |
| | or slow down | N |
| | My breathing makes it difficult to do | 74.5 |
| | things such as walk up hills, carry | |
| | things up | |
| | stairs, light gardening such as | |
| | weeding, dance, play bowls or play | |
| | golf | |
| | My breathing makes it difficult to do | 71.4 |
| | things such as carry heavy loads, dig | |
| | in the garden or shovel snow, jog or | |
| | walk briskly (5 miles per hour), play | |
| | tennis or swim | |
| | My breathing makes it difficult to do | 63.5 |
| | things such as very heavy manual | |
| | work, ride a bike, run, swim fast, or | |
| | play competitive sports | |
| Question 16: We would like to know how | | |
| your respiratory problems usually affect | I cannot play sports or other physical | 64.8 |
| your daily life | activities | w. |
| | I cannot go out for entertainment or | 79.8 |
| | recreation | |
| | I cannot go out of the house to do the | 81.0 |
| | shopping | |
| | I cannot do household chores | 79.1 |
| | I cannot move far from my bed or | 94.0 |
| | chair | |
| Question 17: Tick the statement which | | |
| you think best describes how your | It does not stop me from doing | 0.0 |
| respiratory problems affect you | anything I would like to do | ~ ~~~ |
| | It stops me from doing one or two | 42.0 |
| | things I would like to do | |
| | It stops me from doing most of the | 84.2 |
| | things I would like to do | |





Statistical Analysis Plan 

| It stops me from doing everything I | 96.7 |
|-------------------------------------|------|
| would like to do | |



Statistical Analysis Plan


#### APPENDIX 6. **EQ-5D-5L WEIGHTS**

To account for this study collecting data in multiple countries, different EQ-5D-5L weights will be used depending on the country, as presented in Table 5.

Table 5: EQ-5D-5L geographical region categorisation

| Countries | Version used |
|-------------------------------------------|--------------------------|
| Eastern Europe: Bulgaria, Czech Republic, | Poland (EQ-VT v2.0) |
| Greece, Hungary, Poland, Romania, Russian | 9000 |
| Federation, Slovakia | |
| Western Europe: Germany, United Kingdom | England (EQ-VT v1.0)\ |
| North America: US | US (EQ-VT v2.0) |
| Asia: Republic of Korea | South Korea (EQ-VT v2.0) |

Data collected from questionnaire will be numbered, as presented in Table 6.

Table 6: EQ-5D-5L data collection

| Variable | Mobility | Self- | Usual | Pain/ | Anxiety/ | Health | VAS |
|---|---|---|---|---|---|---|---|
| name | 77.57 | care | Activities | Discomfort | Depression | score | |
| Variable | 1-5 | 1-5 | 1-5 | 1-5 | 1-5 | 5-digit | 0-100 |
| score | | | | | | code for | |
| range | | | | | | EQ-5D-5L | |
| Data row | 2 | 3 | 1 | 1 | 1 | 23111 | 83 |
| example | | | | | | | |

The health score is a combination of the scores for the 5 questions (mobility, self-care, usual activities, pain/discomfort and anxiety/depression) in the order they are collected, as shown in the data row example in Table 6.

#### POLAND

The health index is calculated by first summing all weights related to the scores from the questionnaire and subtracting it from 1, i.e. for data row example in Table 6 the health index would be 0.928. Weights related to each score are presented in Table 7.





Statistical Analysis Plan 

Table 7: Weights

| Variable | Score | Weights |
|---------------------|-------|---------|
| Mobility | 1 | 0 |
| | 2 | 0.025 |
| | 3 | 0.034 |
| | 4 | 0.126 |
| | 5 | 0.314 |
| Self-care | 1 | 0 |
| | 2 | 0.031 |
| | 3 | 0.047 |
| | 4 | 0.111 |
| | 5 | 0.264 |
| Usual Activities | 1 | 0 |
| | 2 | 0.023 |
| | 3 | 0.040 |
| | 4 | 0.097 |
| | 5 | 0.205 |
| Pain/discomfort | 1 | 0 |
| | 2 | 0.030 |
| | 3 | 0.050 |
| | 4 | 0.261 |
| | 5 | 0.575 |
| Anxiety/ depression | 1 | 0 |





Statistical Analysis Plan


| 2 | 0.018 |
|---|-------|
| 3 | 0.029 |
| 4 | 0.108 |
| 5 | 0.232 |

#### ENGLAND

The health index is calculated by first summing all weights related to the scores from the questionnaire and subtracting it from 1, i.e. for data row example in Table 6 the health index would be 0.879. Weights related to each score are presented in Table 8.

Table 8: Weights

| Variable | Score | Weights |
|------------------|-------|---------|
| Mobility | 1 | 0 |
| | 2 | 0.058 |
| | 3 | 0.076 |
| | 4 | 0.207 |
| | 5 | 0.274 |
| Self-care | 1 | 0 |
| | 2 | 0.050 |
| | 3 | 0.080 |
| | 4 | 0.164 |
| | 5 | 0.203 |
| Usual Activities | 1 | 0 |
| | 2 | 0.050 |
| | 3 | 0.063 |





Statistical Analysis Plan


| | 4 | 0.162 |
|---------------------|---|-------|
| | 5 | 0184 |
| Pain/discomfort | 1 | 0 |
| | 2 | 0.063 |
| | 3 | 0.084 |
| | 4 | 0.276 |
| | 5 | 0.335 |
| Anxiety/ depression | 1 | 0 |
| | 2 | 0.078 |
| | 3 | 0.104 |
| | 4 | 0.285 |
| | 5 | 0.289 |

#### US

The health index is calculated by first summing all weights related to the scores from the questionnaire and subtracting it from 1, i.e. for data row example in Table 6 the health index would be 0.797. Weights related to each score are presented in Table 9.

Table 9: Weights

| Variable | Score | Weights |
|----------|-------|---------|
| Mobility | 1 | 0 |
| | 2 | 0.096 |
| | 3 | 0.122 |
| | 4 | 0.237 |
| | 5 | 0.322 |





Statistical Analysis Plan


| Self-care | 1 | 0 |
|---------------------|---|-------|
| | 2 | 0.089 |
| | 3 | 0.107 |
| | 4 | 0.220 |
| | 5 | 0.261 |
| Usual Activities | 1 | 0 |
| | 2 | 0.068 |
| | 3 | 0.101 |
| | 4 | 0.255 |
| | 5 | 0.255 |
| Pain/discomfort | 1 | 0 |
| | 2 | 0.060 |
| | 3 | 0.098 |
| | 4 | 0.318 |
| | 5 | 0.414 |
| Anxiety/ depression | 1 | 0 |
| | 2 | 0.057 |
| | 3 | 0.123 |
| | 4 | 0.299 |
| | 5 | 0.321 |





Statistical Analysis Plan


#### SOUTH KOREA

The value for health state is calculated by first summing all weight related to the score from the questionnaire and subtracting it from 1, i.e. for data row example in Table 6 the value for health state would be 0.875. Weights related to each score are presented in Table 10.

Table 10: Weights

| Variable | Score | Weights |
|---------------------|-------|---------|
| Mobility | 1 | 0 |
| | 2 | 0.063 |
| | 3 | 0.081 |
| | 4 | 0.159 |
| | 5 | 0.268 |
| Self-care | 1 | 0 |
| | 2 | 0.047 |
| | 3 | 0.062 |
| | 4 | 0.095 |
| | 5 | 0.137 |
| Usual Activities | 1 | 0 |
| | 2 | 0.038 |
| | 3 | 0.074 |
| | 4 | 0.127 |
| | 5 | 0.191 |
| Pain/discomfort | 1 | 0 |
| | 2 | 0.052 |
| | 3 | 0.068 |
| | 4 | 0.175 |
| | 5 | 0.226 |
| Anxiety/ depression | 1 | 0 |
| | 2 | 0.042 |
| | 3 | 0.065 |
| | 4 | 0.131 |
| | 5 | 0.157 |



## DocuSign<sup>®</sup>



Electronic Record and Signature Disclosure:

| Payment Events | Status | Timestamps |
|---|---|---|
| Completed | Security Checked | 12/7/2022 5:17:34 AM |
| Envelope Sent Certified Delivered Signing Complete | Hashed/Encrypted Security Checked Security Checked | 12/7/2022 5:16:13 AM<br>12/7/2022 5:17:29 AM<br>12/7/2022 5:17:34 AM |
| Envelope Summary Events | Status | Timestamps 12/6/2022 6:16:13 AM |
| Notary Events | Signature | Timestamp |
| Witness Events | Signature | Timestamp |
| Carbon Copy Events | Status | Timestamp |
| Certified Delivery Events | Status | Timestamp |
| Intermediary Delivery Events | Status | Timestamp |
| Agent Delivery Events | Status | Timestamp |
| Editor Delivery Events | Status | Timestamp |
| In Person Signer Events | Signature | Timestamp |
| Accepted: 12/7/2022 5:17:29 AM ID: a0329438-4184-4e0c-8f5d-0d1ced879e78 Company Name: IQVIA | | |

Signature

Timestamp

Signer Events

**Electronic Record and Signature Disclosure** 

#### CONSENT TO ELECTRONIC DELIVERY AND EXECUTION OF DOCUMENTS

From time to time, IQVIA ("we" or "us") may provide you certain written contracts, notices, disclosures, authorizations, acknowledgements or other documents (collectively, the "Documents") electronically. Please read this consent form carefully. It explains the terms and conditions under which such Documents are provided by us and executed by you electronically through your DocuSign, Inc. ("DocuSign") user account. If you consent to the delivery and execution of such Documents electronically, please click the "I Agree" button.

#### **Documents** will be sent to you electronically

If you consent to electronic delivery, Documents will be sent to your DocuSign user account. You may request a paper copy of documents previously made available through your DocuSign user account, but an additional charge may be incurred. Alternatively, you can download and print documents sent to your DocuSign user account. Unless otherwise noted, you can access a Document up to 30 days from the date we first sent the Document to you.

#### Withhold Consent or Withdrawing Consent to Electronic Delivery

If you withhold consent to electronic delivery or execution, or withdraw your consent at a later date, all Documents will be sent to your mailing address following our receipt of notice of such action. The following sections explain the consequences of withholding or withdrawing your consent to electronic delivery and execution of Documents, and also the procedures you must follow in order to effectuate delivery to your mailing address.

#### **Consequences of Withdrawing Consent**

By electing to only receive and execute Documents sent to your mailing address, we will not be able to carry out transactions or services as efficiently. For instance, some transactions or services require your express consent. We can perform these transaction or services only if we first receive an acknowledgement that indicates you received and consent to the Document related to the proposed transaction or service.

To withhold consent now or withdraw consent at a later date, please sign DocuSign's "Withdraw Consent" form on the signing page of your DocuSign user account. This will indicate that you have withdrawn your consent to receive Documents electronically. Once you sign the "Withdraw Consent" form, you will no longer be able to use your DocuSign user account to execute Documents electronically and we will send Documents to your mailing address. Withdrawal of consent does not affect the validity of any Documents previously executed electronically prior to such withdrawal of Consent. In addition, should you execute any Documents electronically, your execution of such Documents shall indicate your continued consent to execute such Documents electronically.

#### How to contact IQVIA:

If you would like us to send the Documents to a different e-mail address, request paper copies of Documents you have previously received electronically, or withdraw your consent to receive electronic documents, please follow the instructions below. If you have any other questions, please contact: DocuSignSupport@IQVIA.com

#### 1. To advise IQVIA of your new e-mail address

If you would like your Documents sent to a different e-mail address, you must send an e-mail message to DocuSignSupport@IQVIA.com . In the body of the e-mail please state the following: (i) your previous e-mail address, and (ii) your new e-mail address. No other information is required.

In addition, you must notify DocuSign of your new e-mail address. Please log into your DocuSign user account, and follow the instructions to update your e-mail address.

#### 2. To request paper copies from IQVIA

To request paper copies of Documents you have received previously through your DocuSign user account, send an e-mail to DocuSignSupport@IQVIA.com

In the body of the e-mail please state the following: (i) your e-mail address, (ii) full name, (iii) U.S. Postal address, and (iv) telephone number. Additional charges may apply for such paper copies.

#### 3. To withdraw your consent with IQVIA

To withdraw your consent to receiving and executing Documents in an electronic format, you may do one of the following:

i. decline to sign a document from within your DocuSign user account, and on the subsequent page, select the check-box indicating you wish to withdraw your consent; or ii. send us an e-mail to DocuSignSupport@IQVIA.com and in the body of such request you must state your e-mail, full name, US Postal Address, telephone number, and account number. No additional information is necessary.

#### Required hardware and software

| Operating Systems: | Windows® 2000, Windows® XP, Windows Vista®; Mac OS® X |
|---|---|
| Browsers: | <ul> <li>Internet Explorer (Windows Only) 8.0 or above – compatibility mode is supported only for 9.0 and above.</li> <li>Windows Edge Current Version</li> <li>Mozilla Firefox Current Version</li> <li>Safari (Mac OS only) 6.2 or above</li> <li>Google Chrome Current Version</li> </ul> |
| PDF Reader: | Acrobat® or similar software may be required to view and print PDF files |
| Screen Resolution: | 1024 x 768 Recommended |
| Enabled Security Settings: | Allow per session cookies |
| Mobile Signing: | <ul><li>Apple iOS 7.0 or above</li><li>Android 4.0 or above</li></ul> |

<sup>\*\*</sup> These minimum requirements are subject to change. If these requirements change, we will provide you with an e-mail message at the e-mail address we have on file for you at the time the hardware and software requirements are revised.

Pre-release (e.g. beta) versions of operating systems and browsers are not supported.

#### Acknowledging your access and consent to receive materials electronically

To confirm you can access this information electronically and that you consent to receiving and executing Documents electronically on the terms and conditions described above, please let us know by clicking the "I Agree" button.

By clicking the "I Agree" button, you confirm that

- You can access and read this Consent To Electronic Delivery and Execution of Documents; and
- You can print on paper the disclosure or save or send the disclosure to a place where you can print it, for future reference and access; and
- Until or unless you notify IQVIA as described above, you consent to the delivery and execution of Documents electronically.